CLINICAL TRIAL: NCT00996840
Title: Assessment of the Anti-Inflammatory Activity, Efficacy and Safety of Intravenous SB-681323 in Subjects at Risk for Development of Acute Lung Injury (ALI) or Acute Respiratory Distress Syndrome (ARDS).
Brief Title: SB-681323 IV for Subjects at Risk of Acute Lung Injury or ARDS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 111592
Record Dates: First submitted 2009-10-15; First posted 2009-10-16 (Estimated); Results first posted 2017-10-18 (Actual); Last update posted 2017-10-18 (Actual); Status verified 2017-09

CONDITIONS: Lung Injury, Acute
Keywords: dilmapimod; p38; SB-681323; Acute Lung Injury (ALI); Acute Respiratory Distress Syndrome (ARDS)
MeSH Terms: conditions — Acute Lung Injury; Respiratory Distress Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Cohort 1 - SB-681323 Intravenous 3mg (Experimental): 3mg SB-681323 Intravenous administration, infused over 4 hours
  Interventions: Drug: SB-681323 Intravenous 3mg
- Cohort 2 - SB-681323 Intravenous 7.5 mg (Experimental): 7.5 mg SB-681323 Intravenous administration infused over 24 hours
  Interventions: Drug: SB-681323 Intravenous 7.5 mg
- Cohort 3 - SB-681323 Intravenous 7.5mg (Experimental): 7.5 mg SB-681323 Intravenous administration infused over 4 hours
  Interventions: Drug: SB-681323 Intravenous 7.5mg
- Cohort 4 - SB-681323 Intravenous 10mg (Experimental): 10 mg SB-681323 Intravenous administration infused over 24 hours
  Interventions: Drug: SB-681323 Intravenous 10mg
- Combined Placebo (Experimental): Placebo to match intervention
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: SB-681323 Intravenous 3mg — 3 mg SB-681323 Intravenous administration infused over 4 hours
  Arms: Cohort 1 - SB-681323 Intravenous 3mg
Drug: SB-681323 Intravenous 7.5 mg — 7.5 mg SB-681323 Intravenous administration infused over 24 hours
  Arms: Cohort 2 - SB-681323 Intravenous 7.5 mg
Drug: SB-681323 Intravenous 7.5mg — 7.5 mg SB-681323 Intravenous administration infused over 4 hours
  Arms: Cohort 3 - SB-681323 Intravenous 7.5mg
Drug: SB-681323 Intravenous 10mg — 10 mg SB-681323 Intravenous administration infused over 24 hours
  Arms: Cohort 4 - SB-681323 Intravenous 10mg
Other: Placebo — Placebo to match intervention
  Arms: Combined Placebo

SUMMARY:
This is an early phase (Phase IIa), randomized, double-blind, parallel group, multi-centre study for subjects with trauma (physical injury) who are at risk for developing Acute Lung Injury (ALI) or Acute Respiratory Distress Syndrome (ARDS). The primary purpose of the study is to evaluate the safety and tolerability of SB-681323, which is a potent, selective inhibitor of p38 alpha (MAPK) (prevents inflammation of tissue), in comparison to a placebo.

DETAILED DESCRIPTION:
The acute respiratory distress syndrome (ARDS) is a form of severe lung injury (ALI) characterized by hypoxemic respiratory failure (the lungs are unable to absorb oxygen to the arterial blood) and non-cardiogenic pulmonary edema (accumulation of fluid in the lungs). The syndrome may be caused by direct or indirect injury to the lungs. It is associated with a mortality rate of up to 40-50%. There are no marketed pharmacologic therapies for this devastating syndrome.

This study aims to assess the safety and tolerability of SB-681323, which is a potent, selective inhibitor of p38 alpha mitogen-activated protein kinase.

The rationale behind the development of this drug is that there are elevated levels of circulating pro-inflammatory agents, such as cytokines which are biological agents that increase levels of inflammation in the lungs. These agents are part of an 'inflammatory loop' and it may be beneficial to the condition to dampen this loop.

p38 mitogen activated protein kinase (MAPK) plays a major role in the regulation and activation of intracellular proteins which are subsequently involved in the regulation of the cytokines. The pathway is activated by 'stress', such as injury, causing the inflammation. Therefore, 'dampening' this system should reduce the level of inflammation.

This study will investigate the anti-inflammatory activity, efficacy (effectiveness at achieving the desired effect) and safety of SB-681323.

To measure the efficacy of the drug, biomarkers will be measured. Biomarkers are biological agents in the body that are effected by the presence of specific injury or inflammation and are directly or indirectly linked to a regulatory system of event in the body. They are used to measure for the presence and severity of the condition in question. This study will investigate biomarkers linked directly or indirectly to the p38 alpha regulatory mechanism/system. We will be measuring biomarkers such as serum inflammatory biomarkers, coagulation (blood clotting) system biomarkers, biomarkers of endothelial cell / neutrophil interaction and biomarkers of lung epithelial cell injury.

ELIGIBILITY:
Inclusion Criteria:

A subject will be eligible for inclusion in this study only if all of the following criteria apply:

* Male or female, 18 - 80 years of age (inclusive) with major trauma admitted to the Intensive Care Unit (ICU).
* Injury Severity score (ISS) >16 to <70 (exclusive)
* A female subject is eligible to participate if she is of non-child-bearing potential or of:
* Child-bearing potential and agrees to use one of the approved contraception methods (oral contraceptive, either combined or progesterone alone, injectable progesterone, implants of levonorgestrel, estrogenic vaginal ring, percutaneous contraceptive patches, intrauterine device (IUD) or intrauterine system (IUS) with less than 1% non-effectiveness, documented male partner sterilization, double barrier method, i.e. condom and occlusive cap plus spermicidal agent) for an appropriate period of time (as determined by the product label or investigator, if applicable. Female subjects must agree to use contraception until one week post-last dose, if applicable.
* Male subjects must agree to use one of the approved contraception methods (abstinence, defined as sexual inactivity consistent with the preferred and usual lifestyle of the subject, condom during non-vaginal intercourse with any partner (male or female), condom and occlusive cap plus spermicidal agent during sexual intercourse with a female) if applicable. This criterion must be followed from the time of the first dose of study medication until one week post-last dose, if applicable.
* BMI within the range 19.0 - 35.0 kg/m2 inclusive (clinical estimate of height and weight is acceptable).
* The subject or legal decision maker is capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.
* QTcB or QTcF < 450 msec; or QTc < 480 msec in subjects with Bundle Branch Block.
* The subject must be randomized into the study within 24-26 hours from the time of trauma.

Exclusion Criteria:

A subject will not be eligible for inclusion in this study if any of the following criteria apply:

* Known positive Hepatitis B surface antigen or Hepatitis C antibody.
* Known positive test for HIV antibody.
* A known history of substance abuse, alcohol abuse, or regular alcohol consumption within 6 months of the study defined as:
* an average weekly intake of greater than 21 units or an average daily intake of greater than 3 units (males), or defined as an average weekly intake of greater than 14 units or an average daily intake of greater than 2 units (females). One unit is equivalent to a half-pint (220mL) of beer or 1 (25ml) measure of spirits or 1 glass (125ml) of wine.
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* History of sensitivity to any of the study medications, or components thereof, or a history of drug or other allergy that, in the opinion of the investigator or GSK Medical Monitor, contraindicates their participation.
* Haemoglobin < 7g/dL.
* Pregnant females as determined by positive serum or urine hCG test prior to dosing.
* Lactating females.
* Unwillingness or inability to follow the procedures outlined in the protocol.
* History of sensitivity to heparin or heparin-induced thrombocytopenia.
* Diagnosis of ALI at admission.
* Head trauma (Abbreviated Injury Score [AIS]>3), liver trauma (AIS>2), or trauma that in the opinion of the Principle Investigator or GSK medical monitor is deemed unsurvivable.
* Known history of neuromuscular disease or cord injury at C5 or above.
* Elevated ALT or AST > 1.5 ULN.
* History of bone marrow or solid organ transplant.
* Known history of auto-immune disorder in which immunosuppressive agents, other than prednisone, were required within the last 6 weeks.
* Known to be receiving oral or intravenous corticosteroids within 7 days of admission.
* Subject with active tuberculosis or being treated for active tuberculosis.
* Known history of malignancy within the past 5 years with the exception of successfully treated squamous cell or basal cell cancer of the skin.
* Arterial blood pH less than 7.1 or serum HCO3 - <15 before infusion is started.
* Persistent cardiovascular instability requiring therapy with more than one vasopressor.
* A patient will be excluded if in the judgement of the Principle Investigator or GSK medical monitor their participation could jeopardize the health of the subject or the integrity of the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2009-10-16 (Actual); Primary Completion 2013-02-09 (Actual); Study Completion 2013-02-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (6):
- United States (6):
  - GSK Investigational Site, Lexington, Kentucky
  - GSK Investigational Site, Durham, North Carolina
  - GSK Investigational Site, Winston-Salem, North Carolina
  - GSK Investigational Site, Philadelphia, Pennsylvania
  - GSK Investigational Site, Pittsburgh, Pennsylvania
  - GSK Investigational Site, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Christie JD, Vaslef S, Chang PK, May AK, Gunn SR, Yang S, Hardes K, Kahl L, Powley WM, Lipson DA, Bayliffe AI, Lazaar AL. A Randomized Dose-Escalation Study of the Safety and Anti-Inflammatory Activity of the p38 Mitogen-Activated Protein Kinase Inhibitor Dilmapimod in Severe Trauma Subjects at Risk for Acute Respiratory Distress Syndrome. Crit Care Med. 2015 Sep;43(9):1859-69. doi: 10.1097/CCM.0000000000001132. PMID 26102252
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Dataset Specification: 111592 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 111592 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 111592 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 111592 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 111592 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 111592 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 111592 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted across 6 centers in the United States, with 5 centers actually enrolling participants. The first participant was enrolled on 16-October-2009 and the last participant completed the study on 09-February-2013.
Pre-assignment Details: Seventy seven participants were randomized in the study and were included in All subject population.
Groups:
- Combined Placebo: Eligible participants received matching placebo intravenous (IV) infusion over 4 hours (h) or 24 h for 3 days
- Cohort 1-SB-681323, 3 mg, 4 h: Eligible participants received SB-681323, 3 milligrams (mg), IV infusion over 4h for 3 days
- Cohort 2-SB-681323, 7.5 mg, 24 h: Eligible participants received SB-681323, 7.5 mg, IV infusion over 24h for 3 days
- Cohort 3-SB-681323, 7.5 mg, 4 h: Eligible participants received SB-681323, 7.5 mg, IV infusion over 4h for 3 days
- Cohort 4-SB-681323, 10 mg, 24 h: Eligible participants received SB-681323, 10 mg, IV infusion over 24h for 3 days
Period: Overall Study
Arm/Group | Combined Placebo | Cohort 1-SB-681323, 3 mg, 4 h | Cohort 2-SB-681323, 7.5 mg, 24 h | Cohort 3-SB-681323, 7.5 mg, 4 h | Cohort 4-SB-681323, 10 mg, 24 h
Started | 20 | 9 | 12 | 18 | 18
Completed | 19 | 7 | 11 | 17 | 16
Not Completed | 1 | 2 | 1 | 1 | 2
Not completed — Adverse Event | 0 | 1 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 1 | 1 | 2
Not completed — Withdrawal by Subject | 1 | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Combined Placebo: Eligible participants received matching placebo IV infusion over 4 h or 24 h for 3 days
- Cohort 1-SB-681323, 3 mg, 4 h: Eligible participants received SB-681323, 3 mg, IV infusion over 4h for 3 days
- Total: Total of all reporting groups
Arm/Group | Combined Placebo | Cohort 1-SB-681323, 3 mg, 4 h | Cohort 2-SB-681323, 7.5 mg, 24 h | Cohort 3-SB-681323, 7.5 mg, 4 h | Cohort 4-SB-681323, 10 mg, 24 h | Total
Number analyzed (Participants) | 20 | 9 | 12 | 18 | 18 | 77
Age, Continuous [Mean (Standard Deviation); unit: Years] | 41.2 (17.70) | 47.4 (19.31) | 34.5 (15.61) | 44.1 (15.89) | 46.1 (21.80) | 42.7 (18.24)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 1 | 4 | 5 | 16
  Male | 17 | 6 | 11 | 14 | 13 | 61
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 1 | 0 | 1
  Asian | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 8 | 0 | 3 | 3 | 4 | 18
  White | 11 | 9 | 8 | 12 | 13 | 53
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1 | 2 | 1 | 5

OUTCOME MEASURES:

1. Primary Outcome: Mean Hematology Parameters Basophils, Eosinophils, Lymphocytes, Monocytes, Total Neutrophils, Platelet Count, White Blood Cell Count
Description: Mean hematology parameters including basophils, eosinophils, lymphocytes, monocytes, total neutrophils, platelet count, white blood cell count were reported. If sample for hematology test had been obtained for standard of care within ± 4 h of the planned assessment then it was not collected at the planned assessment time point.
Time Frame: "Day 2, pre-dose", "Day 3, pre-dose", "Day 3, 24 h" and "Follow up (Day 7)"
Population: All subject Population comprised of as all participant who received at least one dose of study medication. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Giga cells per liter
Arm/Group | Combined Placebo | Cohort 1-SB-681323, 3 mg, 4 h | Cohort 2-SB-681323, 7.5 mg, 24 h | Cohort 3-SB-681323, 7.5 mg, 4 h | Cohort 4-SB-681323, 10 mg, 24 h
Number analyzed (Participants) | 20 | 9 | 12 | 18 | 18
Giga cells per liter
  Basophils: Day 2, pre-dose: number analyzed (Participants) | 19 | 8 | 12 | 17 | 17
  Basophils: Day 2, pre-dose | 0.0305 (0.04196) | 0.0163 (0.01188) | 0.0208 (0.02843) | 0.0153 (0.01125) | 0.0258 (0.02134)
  Basophils: Day 3, pre-dose: number analyzed (Participants) | 19 | 7 | 11 | 17 | 14
  Basophils: Day 3, pre-dose | 0.0291 (0.03036) | 0.0129 (0.00756) | 0.0209 (0.02737) | 0.0176 (0.01562) | 0.0279 (0.03191)
  Basophils: Day 3, 24 h: number analyzed (Participants) | 18 | 8 | 12 | 17 | 13
  Basophils: Day 3, 24 h | 0.0239 (0.02062) | 0.0294 (0.02809) | 0.0300 (0.02374) | 0.0284 (0.02762) | 0.0315 (0.04240)
  Basophils: Follow up (Day 7): number analyzed (Participants) | 18 | 7 | 10 | 16 | 15
  Basophils: Follow up (Day 7) | 0.0389 (0.03660) | 0.0314 (0.02340) | 0.0300 (0.02625) | 0.0345 (0.03965) | 0.0240 (0.02501)
  Eosinophils: Day 2, pre-dose: number analyzed (Participants) | 19 | 8 | 12 | 17 | 17
  Eosinophils: Day 2, pre-dose | 0.0968 (0.18817) | 0.0676 (0.07149) | 0.0633 (0.07451) | 0.0331 (0.04319) | 0.0724 (0.07411)
  Eosinophils: Day 3, pre-dose: number analyzed (Participants) | 19 | 7 | 11 | 17 | 14
  Eosinophils: Day 3, pre-dose | 0.1588 (0.18027) | 0.0894 (0.06882) | 0.0964 (0.10112) | 0.0746 (0.06376) | 0.0664 (0.04955)
  Eosinophils: Day 3, 24 h: number analyzed (Participants) | 18 | 8 | 12 | 17 | 13
  Eosinophils: Day 3, 24 h | 0.2544 (0.18852) | 0.1538 (0.07558) | 0.1400 (0.14365) | 0.1345 (0.12560) | 0.1142 (0.07005)
  Eosinophils: Follow up (Day 7): number analyzed (Participants) | 19 | 7 | 10 | 16 | 15
  Eosinophils: Follow up (Day 7) | 0.3713 (0.29748) | 0.2866 (0.25120) | 0.1900 (0.16445) | 0.2390 (0.08483) | 0.1998 (0.14855)
  Lymphocytes: Day 2, pre-dose: number analyzed (Participants) | 19 | 8 | 12 | 17 | 17
  Lymphocytes: Day 2, pre-dose | 1.2943 (0.68932) | 0.9725 (0.43980) | 1.0575 (0.49116) | 1.3276 (0.57791) | 1.5365 (0.83119)
  Lymphocytes: Day 3, pre-dose: number analyzed (Participants) | 19 | 7 | 11 | 17 | 14
  Lymphocytes: Day 3, pre-dose | 1.2594 (0.59834) | 1.0103 (0.39949) | 1.0582 (0.42171) | 1.1462 (0.52784) | 1.1593 (0.55383)
  Lymphocytes: Day 3, 24 h: number analyzed (Participants) | 18 | 8 | 12 | 17 | 13
  Lymphocytes: Day 3, 24 h | 1.1146 (0.44206) | 1.0406 (0.36407) | 1.0067 (0.60161) | 1.1936 (0.50190) | 1.4288 (0.62231)
  Lymphocytes: Follow up (Day 7): number analyzed (Participants) | 19 | 7 | 10 | 16 | 15
  Lymphocytes: Follow up (Day 7) | 1.4967 (0.53371) | 1.0611 (0.31455) | 1.0370 (0.50228) | 1.3915 (0.72178) | 1.2835 (0.41700)
  Monocytes: Day 2, pre-dose: number analyzed (Participants) | 19 | 8 | 12 | 17 | 17
  Monocytes: Day 2, pre-dose | 0.8503 (0.36457) | 0.6670 (0.16724) | 0.7900 (0.20432) | 0.9588 (0.53966) | 0.7246 (0.24992)
  Monocytes: Day 3, pre-dose: number analyzed (Participants) | 19 | 7 | 11 | 17 | 14
  Monocytes: Day 3, pre-dose | 0.7726 (0.35421) | 0.6564 (0.20882) | 0.5936 (0.24072) | 0.8479 (0.54882) | 0.6957 (0.22589)
  Monocytes: Day 3, 24 h: number analyzed (Participants) | 18 | 8 | 12 | 17 | 13
  Monocytes: Day 3, 24 h | 0.8554 (0.32384) | 0.6238 (0.16501) | 0.7308 (0.23372) | 0.8852 (0.33731) | 0.6712 (0.29185)
  Monocytes: Follow up (Day 7): number analyzed (Participants) | 19 | 7 | 10 | 16 | 15
  Monocytes: Follow up (Day 7) | 1.1119 (0.50819) | 0.9531 (0.45374) | 0.9030 (0.45314) | 1.1811 (0.42979) | 0.7591 (0.23030)
  Total Neutrophils: Day 2, pre-dose: number analyzed (Participants) | 19 | 8 | 12 | 17 | 17
  Total Neutrophils: Day 2, pre-dose | 9.1607 (2.78517) | 7.0729 (2.28843) | 9.0225 (3.17595) | 9.4199 (2.80762) | 8.2319 (2.78227)
  Total Neutrophils: Day 3, pre-dose: number analyzed (Participants) | 19 | 7 | 11 | 17 | 14
  Total Neutrophils: Day 3, pre-dose | 8.3494 (2.81972) | 6.8724 (2.39872) | 8.6555 (4.16819) | 8.3912 (3.64530) | 8.1779 (2.36852)
  Total Neutrophils: Day 3, 24 h: number analyzed (Participants) | 18 | 8 | 12 | 17 | 13
  Total Neutrophils: Day 3, 24 h | 8.0317 (2.21593) | 5.4550 (2.01330) | 7.7675 (2.93749) | 8.4700 (3.48850) | 6.9604 (3.51501)
  Total Neutrophils: Follow up (Day 7): number analyzed (Participants) | 19 | 7 | 10 | 16 | 15
  Total Neutrophils: Follow up (Day 7) | 9.7596 (3.53180) | 7.8463 (3.49800) | 9.4750 (3.26687) | 9.7576 (4.00884) | 8.4943 (4.71139)
  Platelet count: Day 2, pre-dose: number analyzed (Participants) | 19 | 8 | 12 | 18 | 18
  Platelet count: Day 2, pre-dose | 139.5 (46.84) | 109.6 (36.21) | 152.0 (60.65) | 145.2 (52.96) | 149.5 (45.73)
  Platelet count: Day 3, pre-dose: number analyzed (Participants) | 19 | 8 | 11 | 17 | 17
  Platelet count: Day 3, pre-dose | 143.1 (54.62) | 124.5 (39.16) | 152.4 (66.02) | 144.6 (44.73) | 144.1 (39.33)
  Platelet count: Day 3, 24 h: number analyzed (Participants) | 18 | 8 | 12 | 17 | 17
  Platelet count: Day 3, 24 h | 172.0 (58.25) | 138.9 (28.15) | 177.3 (68.96) | 183.1 (53.62) | 176.1 (44.35)
  Platelet count: Follow up (Day 7): number analyzed (Participants) | 18 | 8 | 12 | 16 | 17
  Platelet count: Follow up (Day 7) | 310.1 (87.28) | 262.4 (76.44) | 253.6 (84.79) | 284.0 (84.37) | 300.6 (105.65)
  White blood cell count: Day 2, pre-dose: number analyzed (Participants) | 20 | 8 | 12 | 18 | 18
  White blood cell count: Day 2, pre-dose | 11.17 (3.394) | 8.80 (2.480) | 10.95 (3.028) | 11.67 (3.377) | 10.88 (3.068)
  White blood cell count: Day 3, pre-dose: number analyzed (Participants) | 20 | 8 | 11 | 17 | 17
  White blood cell count: Day 3, pre-dose | 10.43 (3.482) | 8.55 (2.206) | 10.38 (4.105) | 10.47 (4.112) | 10.36 (2.370)
  White blood cell count: Day 3, 24 h: number analyzed (Participants) | 19 | 8 | 12 | 17 | 17
  White blood cell count: Day 3, 24 h | 10.26 (2.544) | 7.26 (1.859) | 9.68 (2.954) | 10.72 (3.694) | 9.78 (3.316)
  White blood cell count: Follow up (Day 7): number analyzed (Participants) | 19 | 8 | 12 | 17 | 17
  White blood cell count: Follow up (Day 7) | 12.84 (3.894) | 10.73 (3.973) | 11.34 (3.312) | 13.60 (5.614) | 11.18 (5.237)

2. Primary Outcome: Mean Hematology Parameters- Hemoglobin, Mean Corpuscle Hemoglobin Concentration (MCHC)
Description: Mean hematology parameters including hemoglobin, MCHC were reported. If sample for hematology test had been obtained for standard of care within ± 4 h of the planned assessment then it was not collected at the planned assessment time point.
Time Frame: "Day 2, pre-dose", "Day 3, pre-dose", "Day 3, 24 h" and "Follow up (Day 7)"
Population: All subject population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Grams per liter (g/L)
Arm/Group | Combined Placebo | Cohort 1-SB-681323, 3 mg, 4 h | Cohort 2-SB-681323, 7.5 mg, 24 h | Cohort 3-SB-681323, 7.5 mg, 4 h | Cohort 4-SB-681323, 10 mg, 24 h
Number analyzed (Participants) | 20 | 9 | 12 | 18 | 18
Grams per liter (g/L)
  Hemoglobin : Day 2, pre-dose: number analyzed (Participants) | 20 | 8 | 12 | 18 | 18
  Hemoglobin : Day 2, pre-dose | 100.8 (17.05) | 97.0 (16.27) | 97.8 (22.04) | 88.4 (12.46) | 97.2 (20.40)
  Hemoglobin : Day 3, pre-dose: number analyzed (Participants) | 20 | 8 | 11 | 17 | 17
  Hemoglobin : Day 3, pre-dose | 90.6 (15.27) | 96.0 (17.48) | 93.7 (19.40) | 82.9 (9.29) | 95.2 (20.85)
  Hemoglobin : Day 3, 24 h: number analyzed (Participants) | 19 | 8 | 12 | 17 | 17
  Hemoglobin : Day 3, 24 h | 91.9 (12.94) | 96.5 (16.50) | 93.0 (15.36) | 84.7 (9.73) | 95.1 (19.37)
  Hemoglobin: follow up (Day 7): number analyzed (Participants) | 19 | 8 | 12 | 17 | 17
  Hemoglobin: follow up (Day 7) | 94.1 (14.97) | 103.5 (16.42) | 99.6 (15.49) | 88.8 (8.93) | 99.2 (16.36)
  MCHC :Day 2, pre-dose: number analyzed (Participants) | 20 | 8 | 12 | 18 | 18
  MCHC :Day 2, pre-dose | 341.2 (10.96) | 343.8 (4.17) | 339.3 (6.96) | 339.1 (9.43) | 343.6 (10.63)
  MCHC : Day 3, pre-dose: number analyzed (Participants) | 20 | 8 | 11 | 17 | 17
  MCHC : Day 3, pre-dose | 337.4 (9.30) | 343.1 (8.15) | 338.7 (7.64) | 339.1 (7.43) | 341.2 (8.73)
  MCHC : Day 3, 24 h: number analyzed (Participants) | 19 | 8 | 12 | 17 | 17
  MCHC : Day 3, 24 h | 338.2 (9.33) | 342.9 (6.90) | 338.1 (9.34) | 336.4 (10.03) | 342.8 (9.60)
  MCHC : Follow up (Day 7): number analyzed (Participants) | 19 | 8 | 12 | 17 | 17
  MCHC : Follow up (Day 7) | 333.4 (12.09) | 339.5 (10.74) | 337.8 (9.72) | 331.1 (11.89) | 342.5 (9.28)

3. Primary Outcome: Mean Hematology Parameters- Mean Corpuscle Hemoglobin
Description: Hematology parameter mean corpuscle hemoglobin was reported. If sample for hematology test had been obtained for standard of care within ± 4 h of the planned assessment then it was not collected at the planned assessment time point.
Time Frame: "Day 2, pre-dose", "Day 3, pre-dose", "Day 3, 24 h" and "Follow up (Day 7)"
Population: All subject population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Picogram (pg)
Arm/Group | Combined Placebo | Cohort 1-SB-681323, 3 mg, 4 h | Cohort 2-SB-681323, 7.5 mg, 24 h | Cohort 3-SB-681323, 7.5 mg, 4 h | Cohort 4-SB-681323, 10 mg, 24 h
Number analyzed (Participants) | 20 | 9 | 12 | 18 | 18
Picogram (pg)
  Mean Corpuscle Hemoglobin: Day 2, pre-dose: number analyzed (Participants) | 20 | 8 | 12 | 18 | 18
  Mean Corpuscle Hemoglobin: Day 2, pre-dose | 30.46 (1.340) | 30.74 (1.241) | 30.11 (1.262) | 30.18 (1.997) | 31.10 (1.160)
  Mean Corpuscle Hemoglobin: Day 3, pre-dose: number analyzed (Participants) | 20 | 8 | 11 | 17 | 17
  Mean Corpuscle Hemoglobin: Day 3, pre-dose | 30.21 (1.319) | 30.78 (1.290) | 30.22 (1.135) | 30.19 (1.771) | 30.77 (1.332)
  Mean Corpuscle Hemoglobin: Day 3, 24 h: number analyzed (Participants) | 19 | 8 | 12 | 17 | 17
  Mean Corpuscle Hemoglobin: Day 3, 24 h | 30.25 (1.359) | 30.80 (1.153) | 30.33 (1.378) | 30.06 (1.808) | 30.92 (1.274)
  Mean Corpuscle Hemoglobin:Follow up (Day 7): number analyzed (Participants) | 19 | 8 | 12 | 17 | 17
  Mean Corpuscle Hemoglobin:Follow up (Day 7) | 30.02 (1.141) | 30.64 (1.308) | 30.13 (1.234) | 29.82 (1.768) | 31.08 (1.415)

4. Primary Outcome: Hematology Parameters-Mean Corpuscle Volume
Description: Absolute values of mean corpuscle volume were reported. If sample for hematology test had been obtained for standard of care within ± 4 h of the planned assessment then it was not collected at the planned assessment time point.
Time Frame: "Day 2, pre-dose", "Day 3, pre-dose", "Day 3, 24 h" and "Follow up (Day 7)"
Population: All subject population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Femtoliter
Arm/Group | Combined Placebo | Cohort 1-SB-681323, 3 mg, 4 h | Cohort 2-SB-681323, 7.5 mg, 24 h | Cohort 3-SB-681323, 7.5 mg, 4 h | Cohort 4-SB-681323, 10 mg, 24 h
Number analyzed (Participants) | 20 | 9 | 12 | 18 | 18
Femtoliter
  Mean Corpuscle Volume:Day 2, pre-dose: number analyzed (Participants) | 20 | 8 | 12 | 18 | 18
  Mean Corpuscle Volume:Day 2, pre-dose | 89.30 (4.024) | 89.59 (3.379) | 88.33 (3.367) | 89.15 (4.828) | 90.63 (2.809)
  Mean Corpuscle Volume: Day 3, pre-dose: number analyzed (Participants) | 20 | 8 | 11 | 17 | 17
  Mean Corpuscle Volume: Day 3, pre-dose | 89.85 (3.833) | 89.70 (2.804) | 89.00 (3.742) | 89.18 (4.375) | 90.48 (3.075)
  Mean Corpuscle Volume: Day 3, 24 h: number analyzed (Participants) | 19 | 8 | 12 | 17 | 17
  Mean Corpuscle Volume: Day 3, 24 h | 89.41 (3.920) | 89.96 (2.295) | 89.50 (3.920) | 89.45 (4.285) | 90.08 (2.510)
  Mean Corpuscle Volume: Follow up (Day 7): number analyzed (Participants) | 19 | 8 | 12 | 17 | 17
  Mean Corpuscle Volume: Follow up (Day 7) | 90.12 (3.430) | 89.86 (2.738) | 89.67 (3.869) | 90.43 (4.079) | 90.75 (3.115)

5. Primary Outcome: Mean Hematology Parameters-reticulocytes, Red Blood Cell Count
Description: Absolute values of reticulocytes and red blood cell count were reported. If sample for hematology test had been obtained for standard of care within ± 4 h of the planned assessment then it was not collected at the planned assessment time point.
Time Frame: "Day 2, pre-dose", "Day 3, pre-dose", "Day 3, 24 h" and "Follow up (Day 7)"
Population: All subject population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Trillion cells per liter (TI/L)
Arm/Group | Combined Placebo | Cohort 1-SB-681323, 3 mg, 4 h | Cohort 2-SB-681323, 7.5 mg, 24 h | Cohort 3-SB-681323, 7.5 mg, 4 h | Cohort 4-SB-681323, 10 mg, 24 h
Number analyzed (Participants) | 20 | 9 | 12 | 18 | 18
Trillion cells per liter (TI/L)
  Reticulocytes : Day 2, pre-dose: number analyzed (Participants) | 19 | 7 | 12 | 16 | 15
  Reticulocytes : Day 2, pre-dose | 0.0488 (0.01974) | 0.0411 (0.01902) | 0.0406 (0.00863) | 0.0398 (0.01218) | 0.0513 (0.02192)
  Reticulocytes : Day 3, pre-dose: number analyzed (Participants) | 20 | 8 | 11 | 17 | 12
  Reticulocytes : Day 3, pre-dose | 0.0554 (0.01871) | 0.0448 (0.01903) | 0.0464 (0.01284) | 0.0474 (0.01382) | 0.0576 (0.02543)
  Reticulocytes : Day 3, 24 h: number analyzed (Participants) | 18 | 7 | 12 | 17 | 13
  Reticulocytes : Day 3, 24 h | 0.0662 (0.02171) | 0.0592 (0.02654) | 0.0538 (0.01876) | 0.0581 (0.01748) | 0.0699 (0.02818)
  Reticulocytes : Follow up (Day 7): number analyzed (Participants) | 17 | 8 | 9 | 17 | 13
  Reticulocytes : Follow up (Day 7) | 0.0934 (0.04509) | 0.0979 (0.04134) | 0.0829 (0.05170) | 0.0897 (0.03964) | 0.1213 (0.06734)
  Red Blood Cell count : Day 2, pre-dose: number analyzed (Participants) | 20 | 8 | 12 | 18 | 18
  Red Blood Cell count : Day 2, pre-dose | 3.320 (0.6164) | 3.151 (0.4434) | 3.253 (0.6883) | 2.943 (0.4695) | 3.121 (0.6197)
  Red Blood Cell count : Day 3, pre-dose: number analyzed (Participants) | 20 | 8 | 11 | 17 | 17
  Red Blood Cell count : Day 3, pre-dose | 3.007 (0.5787) | 3.110 (0.5001) | 3.103 (0.6117) | 2.758 (0.3615) | 3.083 (0.6114)
  Red Blood Cell count : Day 3, 24 h: number analyzed (Participants) | 19 | 8 | 12 | 17 | 17
  Red Blood Cell count : Day 3, 24 h | 3.054 (0.5220) | 3.128 (0.4706) | 3.071 (0.5146) | 2.822 (0.3372) | 3.062 (0.5799)
  Red Blood Cell count : Follow up (Day 7): number analyzed (Participants) | 19 | 8 | 12 | 17 | 17
  Red Blood Cell count : Follow up (Day 7) | 3.144 (0.5268) | 3.379 (0.4695) | 3.313 (0.5365) | 2.983 (0.3445) | 3.183 (0.4403)

6. Primary Outcome: Mean Clinical Chemistry Parameters- Albumin and Total Protein
Description: Absolute values of albumin and total protein were reported. If sample for clinical chemistry test had been obtained for standard of care within ± 4 h of the planned assessment then it was not collected at the planned assessment time point.
Time Frame: "Day 2, pre-dose", "Day 3, pre-dose", "Day 3, 24 h" and "Follow up (Day 7)"
Population: All subject population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Combined Placebo | Cohort 1-SB-681323, 3 mg, 4 h | Cohort 2-SB-681323, 7.5 mg, 24 h | Cohort 3-SB-681323, 7.5 mg, 4 h | Cohort 4-SB-681323, 10 mg, 24 h
Number analyzed (Participants) | 20 | 9 | 12 | 18 | 18
g/L
  Albumin : Day 2, pre-dose: number analyzed (Participants) | 20 | 8 | 11 | 18 | 15
  Albumin : Day 2, pre-dose | 25.2 (4.27) | 25.1 (5.72) | 23.7 (3.69) | 26.2 (3.45) | 24.7 (5.33)
  Albumin : Day 3, pre-dose: number analyzed (Participants) | 20 | 8 | 11 | 17 | 15
  Albumin : Day 3, pre-dose | 22.8 (4.29) | 25.6 (4.96) | 22.6 (5.45) | 23.1 (3.51) | 25.1 (6.06)
  Albumin : Day 3, 24 h: number analyzed (Participants) | 19 | 7 | 12 | 17 | 13
  Albumin : Day 3, 24 h | 22.4 (3.99) | 24.1 (4.56) | 22.7 (4.85) | 22.6 (3.90) | 24.3 (6.69)
  Albumin : Follow up (Day 7): number analyzed (Participants) | 18 | 8 | 10 | 17 | 14
  Albumin : Follow up (Day 7) | 22.4 (6.34) | 25.5 (4.87) | 21.6 (4.74) | 22.0 (3.86) | 26.8 (5.03)
  Total Protein : Day 2, pre-dose: number analyzed (Participants) | 20 | 7 | 11 | 16 | 16
  Total Protein : Day 2, pre-dose | 49.4 (7.39) | 47.1 (9.44) | 46.8 (7.64) | 48.9 (5.76) | 51.1 (9.21)
  Total Protein : Day 3, pre-dose: number analyzed (Participants) | 20 | 7 | 10 | 17 | 16
  Total Protein : Day 3, pre-dose | 47.8 (8.01) | 50.0 (7.02) | 46.3 (9.24) | 47.1 (3.82) | 52.7 (11.24)
  Total Protein : Day 3, 24 h: number analyzed (Participants) | 19 | 7 | 11 | 17 | 14
  Total Protein : Day 3, 24 h | 51.4 (7.09) | 49.6 (3.82) | 49.2 (7.78) | 49.0 (5.00) | 53.2 (10.99)
  Total Protein : Follow up (Day 7): number analyzed (Participants) | 18 | 8 | 9 | 17 | 14
  Total Protein : Follow up (Day 7) | 55.8 (9.54) | 55.6 (4.27) | 50.3 (8.66) | 52.3 (7.41) | 58.5 (8.55)

7. Primary Outcome: Mean Clinical Chemistry Parameters-alkaline Phosphatase, Alanine Amino Transferase, Aspartate Amino Transferase, Creatine Kinase and Gamma Glutamyl Transferase
Description: Absolute values of alkaline phosphatase, alanine amino transferase, aspartate amino transferase, creatine kinase and gamma glutamyl transferase were reported. If sample for clinical chemistry test had been obtained for standard of care within ± 4 h of the planned assessment then it was not collected at the planned assessment time point.
Time Frame: "Day 2, pre-dose", "Day 3, pre-dose", "Day 3, 24 h" and "Follow up (Day 7)"
Population: All subject population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: International units per liter (IU/L)
Arm/Group | Combined Placebo | Cohort 1-SB-681323, 3 mg, 4 h | Cohort 2-SB-681323, 7.5 mg, 24 h | Cohort 3-SB-681323, 7.5 mg, 4 h | Cohort 4-SB-681323, 10 mg, 24 h
Number analyzed (Participants) | 20 | 9 | 12 | 18 | 18
International units per liter (IU/L)
  Alkaline phosphatase : Day 2, pre-dose: number analyzed (Participants) | 20 | 8 | 11 | 18 | 18
  Alkaline phosphatase : Day 2, pre-dose | 52.0 (19.99) | 53.8 (12.53) | 43.5 (8.19) | 49.4 (21.15) | 52.2 (17.98)
  Alkaline phosphatase : Day 3, pre-dose: number analyzed (Participants) | 20 | 8 | 11 | 17 | 16
  Alkaline phosphatase : Day 3, pre-dose | 52.6 (20.35) | 73.1 (45.57) | 48.6 (11.07) | 50.8 (26.85) | 55.6 (18.92)
  Alkaline phosphatase : Day 3, 24 h: number analyzed (Participants) | 19 | 8 | 11 | 17 | 15
  Alkaline phosphatase : Day 3, 24 h | 66.6 (37.08) | 76.0 (44.67) | 53.5 (13.19) | 60.6 (34.38) | 59.5 (25.61)
  Alkaline phosphatase : Follow up (Day 7): number analyzed (Participants) | 19 | 8 | 9 | 17 | 16
  Alkaline phosphatase : Follow up (Day 7) | 89.3 (57.58) | 118.1 (58.77) | 69.8 (39.40) | 94.5 (59.93) | 90.0 (60.86)
  Alanine Amino Transferase : Day 2, pre-dose: number analyzed (Participants) | 20 | 8 | 11 | 18 | 18
  Alanine Amino Transferase : Day 2, pre-dose | 51.1 (26.48) | 37.8 (26.63) | 60.5 (37.89) | 45.4 (22.67) | 53.8 (49.17)
  Alanine Amino Transferase : Day 3, pre-dose: number analyzed (Participants) | 20 | 8 | 11 | 17 | 16
  Alanine Amino Transferase : Day 3, pre-dose | 43.1 (18.64) | 43.4 (48.84) | 50.8 (26.93) | 37.5 (15.91) | 41.4 (32.89)
  Alanine Amino Transferase : Day 3, 24 h: number analyzed (Participants) | 19 | 8 | 11 | 17 | 16
  Alanine Amino Transferase : Day 3, 24 h | 44.7 (21.93) | 53.3 (62.19) | 49.1 (21.82) | 34.3 (15.14) | 42.3 (29.56)
  Alanine Amino Transferase : Follow up (Day 7): number analyzed (Participants) | 19 | 8 | 9 | 17 | 16
  Alanine Amino Transferase : Follow up (Day 7) | 52.5 (50.95) | 77.4 (58.39) | 117.8 (158.33) | 42.2 (21.73) | 59.1 (52.41)
  Aspartate Amino Transferase : Day 2, pre-dose: number analyzed (Participants) | 20 | 8 | 11 | 18 | 18
  Aspartate Amino Transferase : Day 2, pre-dose | 74.6 (42.35) | 57.1 (28.41) | 125.2 (65.22) | 83.2 (40.61) | 81.4 (53.72)
  Aspartate Amino Transferase : Day 3, pre-dose: number analyzed (Participants) | 20 | 8 | 11 | 17 | 16
  Aspartate Amino Transferase : Day 3, pre-dose | 73.3 (62.80) | 64.9 (58.77) | 90.5 (44.66) | 65.8 (31.23) | 62.3 (29.70)
  Aspartate Amino Transferase : Day 3, 24 h: number analyzed (Participants) | 19 | 8 | 11 | 17 | 16
  Aspartate Amino Transferase : Day 3, 24 h | 77.5 (93.43) | 81.3 (79.91) | 84.9 (37.84) | 53.1 (29.14) | 71.9 (66.70)
  Aspartate Amino Transferase : Follow up (Day 7): number analyzed (Participants) | 19 | 8 | 9 | 17 | 16
  Aspartate Amino Transferase : Follow up (Day 7) | 57.9 (46.83) | 64.9 (31.73) | 137.1 (192.21) | 48.3 (21.76) | 65.6 (59.80)
  Creatine Kinase : Day 2, pre-dose: number analyzed (Participants) | 19 | 8 | 11 | 17 | 17
  Creatine Kinase : Day 2, pre-dose | 3287.8 (3333.83) | 1174.0 (996.71) | 4663.1 (4797.79) | 2797.2 (2022.44) | 2527.8 (2507.94)
  Creatine Kinase : Day 3, pre-dose: number analyzed (Participants) | 20 | 8 | 11 | 17 | 17
  Creatine Kinase : Day 3, pre-dose | 2668.0 (4149.97) | 1183.8 (944.80) | 4418.9 (5201.64) | 2307.0 (1670.81) | 2418.9 (3267.70)
  Creatine Kinase : Day 3, 24 h: number analyzed (Participants) | 19 | 7 | 12 | 17 | 13
  Creatine Kinase : Day 3, 24 h | 2527.4 (5594.82) | 1638.3 (2178.26) | 3342.3 (2222.65) | 1410.2 (1417.50) | 1227.8 (1038.81)
  Creatine Kinase : Follow up (Day 7): number analyzed (Participants) | 18 | 8 | 9 | 17 | 15
  Creatine Kinase : Follow up (Day 7) | 954.3 (2023.51) | 503.8 (725.49) | 1349.9 (1296.97) | 602.1 (476.66) | 366.4 (329.52)
  Gamma Glutamyl Transferase : Day 2, pre-dose: number analyzed (Participants) | 20 | 8 | 11 | 17 | 17
  Gamma Glutamyl Transferase : Day 2, pre-dose | 25.2 (20.05) | 20.8 (8.80) | 34.0 (46.54) | 26.3 (23.01) | 17.3 (11.67)
  Gamma Glutamyl Transferase : Day 3, pre-dose: number analyzed (Participants) | 20 | 8 | 11 | 16 | 15
  Gamma Glutamyl Transferase : Day 3, pre-dose | 27.3 (23.02) | 23.0 (9.81) | 25.4 (15.36) | 23.7 (18.42) | 26.9 (31.60)
  Gamma Glutamyl Transferase : Day 3, 24 h: number analyzed (Participants) | 19 | 8 | 11 | 16 | 13
  Gamma Glutamyl Transferase : Day 3, 24 h | 39.4 (47.61) | 31.3 (22.68) | 38.4 (33.91) | 43.4 (46.70) | 39.3 (54.64)
  Gamma Glutamyl Transferase : Follow up (Day 7): number analyzed (Participants) | 18 | 8 | 9 | 17 | 14
  Gamma Glutamyl Transferase : Follow up (Day 7) | 75.9 (61.62) | 70.6 (49.58) | 48.3 (41.93) | 86.7 (90.58) | 45.6 (46.01)

8. Primary Outcome: Mean Clinical Chemistry Parameters- Direct Bilirubin, Total Bilirubin, Creatinine and Uric Acid
Description: Absolute values of direct bilirubin, total bilirubin, creatinine and uric acid were reported. If sample for clinical chemistry test had been obtained for standard of care within ± 4 h of the planned assessment then it was not collected at the planned assessment time point.
Time Frame: "Day 2, pre-dose", "Day 3, pre-dose", "Day 3, 24 h" and "Follow up (Day 7)"
Population: All subject population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Micromol per liter
Arm/Group | Combined Placebo | Cohort 1-SB-681323, 3 mg, 4 h | Cohort 2-SB-681323, 7.5 mg, 24 h | Cohort 3-SB-681323, 7.5 mg, 4 h | Cohort 4-SB-681323, 10 mg, 24 h
Number analyzed (Participants) | 20 | 9 | 12 | 18 | 18
Micromol per liter
  Direct Bilirubin : Day 2, pre-dose: number analyzed (Participants) | 19 | 8 | 11 | 16 | 15
  Direct Bilirubin : Day 2, pre-dose | 4.500 (1.6333) | 4.275 (2.0438) | 8.705 (11.6846) | 5.985 (6.9250) | 3.306 (1.6436)
  Direct Bilirubin : Day 3, pre-dose: number analyzed (Participants) | 19 | 8 | 11 | 17 | 13
  Direct Bilirubin : Day 3, pre-dose | 4.590 (1.9789) | 4.275 (1.5832) | 6.995 (7.2329) | 6.840 (9.5974) | 3.420 (2.2076)
  Direct Bilirubin : Day 3, 24 h: number analyzed (Participants) | 18 | 8 | 11 | 17 | 13
  Direct Bilirubin : Day 3, 24 h | 5.890 (4.0305) | 4.703 (2.5446) | 7.773 (10.6340) | 6.639 (9.7463) | 4.998 (4.1572)
  Direct Bilirubin : Follow up (Day 7): number analyzed (Participants) | 19 | 8 | 9 | 17 | 15
  Direct Bilirubin : Follow up (Day 7) | 7.110 (5.7923) | 7.695 (8.7671) | 26.030 (58.4146) | 10.964 (22.2140) | 9.120 (16.4864)
  Total Bilirubin : Day 2, pre-dose: number analyzed (Participants) | 20 | 8 | 11 | 18 | 18
  Total Bilirubin : Day 2, pre-dose | 19.238 (9.9071) | 17.314 (8.7403) | 24.717 (16.4971) | 15.675 (8.8223) | 18.145 (14.8048)
  Total Bilirubin : Day 3, pre-dose: number analyzed (Participants) | 20 | 8 | 11 | 17 | 16
  Total Bilirubin : Day 3, pre-dose | 18.126 (6.1128) | 16.245 (5.9937) | 20.520 (14.7497) | 18.408 (11.8245) | 15.604 (6.7214)
  Total Bilirubin : Day 3, 24 h: number analyzed (Participants) | 19 | 8 | 11 | 17 | 16
  Total Bilirubin : Day 3, 24 h | 20.430 (7.6574) | 19.238 (8.1112) | 21.608 (15.0494) | 19.615 (12.2882) | 18.596 (9.6505)
  Total Bilirubin : Follow up (Day 7): number analyzed (Participants) | 19 | 8 | 9 | 17 | 16
  Total Bilirubin : Follow up (Day 7) | 20.880 (8.4271) | 24.581 (15.2383) | 53.390 (98.8728) | 26.656 (30.4820) | 22.978 (22.7112)
  Creatinine : Day 2, pre-dose: number analyzed (Participants) | 20 | 8 | 11 | 18 | 18
  Creatinine : Day 2, pre-dose | 76.6428 (23.25282) | 83.4275 (49.48807) | 87.9982 (34.95181) | 90.9538 (66.75768) | 80.1984 (32.87944)
  Creatinine : Day 3, pre-dose: number analyzed (Participants) | 20 | 8 | 11 | 17 | 17
  Creatinine : Day 3, pre-dose | 71.1620 (22.69678) | 80.2230 (51.77845) | 87.9178 (53.40174) | 87.4640 (65.10727) | 72.9560 (31.73042)
  Creatinine : Day 3, 24 h: number analyzed (Participants) | 19 | 8 | 12 | 17 | 16
  Creatinine : Day 3, 24 h | 69.9756 (22.20243) | 73.0405 (45.07022) | 89.7260 (84.44314) | 90.8960 (91.11701) | 78.1788 (28.17353)
  Creatinine : Follow up (Day 7): number analyzed (Participants) | 19 | 8 | 12 | 17 | 17
  Creatinine : Follow up (Day 7) | 70.7200 (25.41831) | 71.8250 (31.43842) | 85.9690 (61.38913) | 98.7480 (110.4008) | 76.9080 (35.07431)
  Uric acid : Day 2, pre-dose: number analyzed (Participants) | 20 | 8 | 11 | 18 | 16
  Uric acid : Day 2, pre-dose | 200.7450 (79.77454) | 207.4365 (76.26689) | 194.1211 (99.68084) | 246.5116 (96.00019) | 231.9720 (76.04761)
  Uric acid : Day 3, pre-dose: number analyzed (Participants) | 20 | 8 | 11 | 17 | 15
  Uric acid : Day 3, pre-dose | 185.2802 (76.68988) | 202.9755 (83.29855) | 202.7727 (83.20631) | 233.3715 (101.8900) | 226.4205 (79.05205)
  Uric acid : Day 3, 24 h: number analyzed (Participants) | 19 | 8 | 11 | 17 | 15
  Uric acid : Day 3, 24 h | 190.6491 (75.69201) | 194.0535 (90.48210) | 192.4989 (95.58615) | 222.8751 (115.7210) | 247.0403 (87.73096)
  Uric acid : Follow up (Day 7): number analyzed (Participants) | 18 | 8 | 8 | 17 | 15
  Uric acid : Follow up (Day 7) | 174.4747 (74.95979) | 171.0050 (62.36289) | 188.8490 (106.1990) | 221.4755 (129.6427) | 253.7813 (118.3352)

9. Primary Outcome: Mean Clinical Chemistry Parameters- Calcium, Chloride, Glucose, Bicarbonate, Potassium, Sodium and Ratio of Urea to Blood Urea Nitrogen (Urea/BUN)
Description: Absolute values of calcium, chloride, glucose, bicarbonate, potassium, sodium and Urea/BUN were reported. If sample for clinical chemistry test had been obtained for standard of care within ± 4 h of the planned assessment then it was not collected at the planned assessment time point.
Time Frame: "Day 2, pre-dose", "Day 3, pre-dose", "Day 3, 24 h" and "Follow up (Day 7)"
Population: All subject population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Millimole per liter
Arm/Group | Combined Placebo | Cohort 1-SB-681323, 3 mg, 4 h | Cohort 2-SB-681323, 7.5 mg, 24 h | Cohort 3-SB-681323, 7.5 mg, 4 h | Cohort 4-SB-681323, 10 mg, 24 h
Number analyzed (Participants) | 20 | 9 | 12 | 18 | 18
Millimole per liter
  Calcium : Day 2, pre-dose: number analyzed (Participants) | 20 | 8 | 11 | 18 | 18
  Calcium : Day 2, pre-dose | 1.9523 (0.11501) | 1.9274 (0.12913) | 1.9098 (0.11828) | 1.9489 (0.08889) | 1.9655 (0.13867)
  Calcium : Day 3, pre-dose: number analyzed (Participants) | 20 | 8 | 11 | 17 | 17
  Calcium : Day 3, pre-dose | 1.9523 (0.10857) | 1.9835 (0.11158) | 1.9007 (0.08411) | 1.9314 (0.12383) | 1.9887 (0.15273)
  Calcium : Day 3, 24 h: number analyzed (Participants) | 19 | 8 | 12 | 17 | 16
  Calcium : Day 3, 24 h | 1.9881 (0.09701) | 2.0272 (0.09312) | 1.9565 (0.15138) | 1.9432 (0.09120) | 2.0116 (0.15132)
  Calcium : Follow up (Day 7): number analyzed (Participants) | 19 | 8 | 11 | 17 | 17
  Calcium : Follow up (Day 7) | 2.0617 (0.14021) | 2.0989 (0.12612) | 2.0005 (0.15773) | 2.0386 (0.11794) | 2.0958 (0.14441)
  Chloride : Day 2, pre-dose: number analyzed (Participants) | 20 | 8 | 11 | 18 | 18
  Chloride : Day 2, pre-dose | 106.5 (5.04) | 105.5 (4.69) | 107.5 (3.62) | 106.3 (4.17) | 105.3 (4.75)
  Chloride : Day 3, pre-dose: number analyzed (Participants) | 20 | 8 | 11 | 17 | 17
  Chloride : Day 3, pre-dose | 106.3 (5.66) | 105.5 (4.93) | 107.7 (4.67) | 105.9 (5.89) | 105.7 (4.25)
  Chloride : Day 3, 24 h: number analyzed (Participants) | 19 | 8 | 12 | 17 | 16
  Chloride : Day 3, 24 h | 104.6 (5.12) | 104.4 (4.98) | 106.0 (5.54) | 106.4 (5.84) | 105.3 (4.41)
  Chloride : Follow up (Day 7): number analyzed (Participants) | 19 | 8 | 11 | 17 | 17
  Chloride : Follow up (Day 7) | 105.2 (7.84) | 101.8 (4.59) | 106.2 (5.13) | 104.5 (6.07) | 102.2 (3.15)
  Glucose : Day 2, pre-dose: number analyzed (Participants) | 20 | 8 | 11 | 18 | 18
  Glucose : Day 2, pre-dose | 6.8028 (2.22918) | 8.0628 (1.92721) | 6.9690 (1.03682) | 7.8763 (2.30585) | 7.3797 (4.08342)
  Glucose : Day 3, pre-dose: number analyzed (Participants) | 20 | 8 | 11 | 17 | 17
  Glucose : Day 3, pre-dose | 6.7889 (1.93504) | 7.2094 (1.67306) | 6.2878 (1.22124) | 7.8530 (2.96473) | 6.2530 (0.98343)
  Glucose : Day 3, 24 h: number analyzed (Participants) | 19 | 8 | 12 | 17 | 15
  Glucose : Day 3, 24 h | 7.6575 (4.44567) | 6.2865 (1.01307) | 6.1662 (0.84863) | 7.7192 (3.27506) | 6.0321 (1.32273)
  Glucose : Follow up (Day 7): number analyzed (Participants) | 19 | 8 | 11 | 16 | 17
  Glucose : Follow up (Day 7) | 6.6115 (1.95391) | 6.3698 (0.55172) | 6.4139 (1.50295) | 6.9110 (2.14454) | 6.2563 (1.41547)
  Bicarbonate : Day 2, pre-dose: number analyzed (Participants) | 20 | 9 | 11 | 18 | 18
  Bicarbonate : Day 2, pre-dose | 26.0 (2.73) | 25.9 (2.36) | 25.6 (2.11) | 25.9 (2.55) | 25.6 (2.20)
  Bicarbonate : Day 3, pre-dose: number analyzed (Participants) | 20 | 9 | 11 | 17 | 17
  Bicarbonate : Day 3, pre-dose | 27.2 (1.96) | 27.8 (2.92) | 26.5 (2.91) | 26.5 (3.47) | 25.7 (2.69)
  Bicarbonate : Day 3, 24 h: number analyzed (Participants) | 19 | 9 | 12 | 17 | 16
  Bicarbonate : Day 3, 24 h | 27.7 (2.70) | 28.5 (2.62) | 27.3 (3.86) | 26.6 (2.18) | 25.3 (2.59)
  Bicarbonate : Follow up (Day 7): number analyzed (Participants) | 19 | 9 | 12 | 17 | 17
  Bicarbonate : Follow up (Day 7) | 27.3 (2.75) | 27.3 (2.49) | 28.3 (1.91) | 27.1 (2.67) | 26.7 (3.14)
  Potassium : Day 2, pre-dose: number analyzed (Participants) | 20 | 8 | 11 | 18 | 18
  Potassium : Day 2, pre-dose | 4.22 (0.558) | 3.89 (0.348) | 4.17 (0.374) | 4.10 (0.468) | 4.12 (0.342)
  Potassium : Day 3, pre-dose: number analyzed (Participants) | 20 | 8 | 11 | 17 | 17
  Potassium : Day 3, pre-dose | 3.88 (0.318) | 3.96 (0.267) | 4.15 (0.491) | 4.00 (0.550) | 3.99 (0.376)
  Potassium : Day 3, 24 h: number analyzed (Participants) | 19 | 8 | 12 | 17 | 15
  Potassium : Day 3, 24 h | 3.85 (0.347) | 3.91 (0.280) | 3.93 (0.442) | 3.91 (0.496) | 3.95 (0.449)
  Potassium : Follow up (Day 7): number analyzed (Participants) | 19 | 8 | 12 | 17 | 17
  Potassium : Follow up (Day 7) | 4.01 (0.435) | 4.01 (0.473) | 3.70 (0.357) | 3.99 (0.405) | 3.98 (0.256)
  Sodium : Day 2, pre-dose: number analyzed (Participants) | 20 | 8 | 11 | 18 | 18
  Sodium : Day 2, pre-dose | 137.1 (3.61) | 136.3 (3.45) | 136.7 (3.44) | 136.7 (2.97) | 137.2 (4.02)
  Sodium : Day 3, pre-dose: number analyzed (Participants) | 20 | 8 | 11 | 17 | 17
  Sodium : Day 3, pre-dose | 138.0 (3.91) | 138.4 (3.29) | 138.5 (3.80) | 137.6 (3.69) | 138.1 (3.66)
  Sodium : Day 3, 24 h: number analyzed (Participants) | 19 | 8 | 12 | 17 | 16
  Sodium : Day 3, 24 h | 138.2 (4.15) | 137.9 (3.48) | 138.5 (3.09) | 138.4 (3.86) | 137.9 (3.24)
  Sodium : Follow up (Day 7): number analyzed (Participants) | 19 | 8 | 12 | 17 | 17
  Sodium : Follow up (Day 7) | 139.6 (5.96) | 137.1 (4.97) | 140.2 (5.22) | 139.0 (5.05) | 136.6 (3.06)
  Urea/BUN : Day 2, pre-dose: number analyzed (Participants) | 20 | 8 | 11 | 18 | 18
  Urea/BUN : Day 2, pre-dose | 3.7664 (2.13093) | 3.4361 (3.16986) | 4.3392 (3.00056) | 4.9385 (3.44877) | 4.6013 (2.85045)
  Urea/BUN : Day 3, pre-dose: number analyzed (Participants) | 20 | 8 | 11 | 17 | 17
  Urea/BUN : Day 3, pre-dose | 3.4808 (1.57061) | 3.7485 (3.85447) | 4.9655 (4.52265) | 4.8510 (3.92306) | 4.6200 (2.93162)
  Urea/BUN : Day 3, 24 h: number analyzed (Participants) | 19 | 8 | 12 | 17 | 16
  Urea/BUN : Day 3, 24 h | 4.1525 (2.34164) | 4.3286 (4.26883) | 4.9683 (6.06128) | 5.4390 (5.13095) | 4.8418 (2.59399)
  Urea/BUN : Follow up (Day 7): number analyzed (Participants) | 19 | 8 | 11 | 17 | 17
  Urea/BUN : Follow up (Day 7) | 5.9938 (5.08449) | 6.0244 (4.20870) | 6.2313 (7.18868) | 7.1610 (8.27331) | 5.3340 (2.80100)

10. Primary Outcome: Mean Clinical Chemistry Parameters-estradiol
Description: Absolute values of Estradiol were reported. If sample for clinical chemistry test had been obtained for standard of care within ± 4 h of the planned assessment then it was not collected at the planned assessment time point.
Time Frame: Day 1 (pre-dose) and Day 3 (24 h)
Population: All subject population. Only those participants available at the specified time points were analyzed. Data were not collected from participants in Cohort 2-SB-681323, 7.5 mg, 24 h, Cohort 3-SB-681323, 7.5 mg, 4 h, and Cohort 4-SB-681323, 10 mg, 24 h.
Measure: Mean (Standard Deviation); unit: Picomole per liter
Arm/Group | Combined Placebo | Cohort 1-SB-681323, 3 mg, 4 h | Cohort 2-SB-681323, 7.5 mg, 24 h | Cohort 3-SB-681323, 7.5 mg, 4 h | Cohort 4-SB-681323, 10 mg, 24 h
Number analyzed (Participants) | 1 | 4 | 0 | 0 | 0
Picomole per liter | 165.150 (NA) — Only one participant was available at the time of analysis, dispersion could not be calculated. | 210.108 (100.8360) |  |  |

11. Primary Outcome: Mean Clinical Chemistry Parameters-Blood pH at Screening
Description: Absolute values of Blood pH at screening were reported as clinical chemistry parameter.
Time Frame: Screening
Population: All subject population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: pH Units
Arm/Group | Combined Placebo | Cohort 1-SB-681323, 3 mg, 4 h | Cohort 2-SB-681323, 7.5 mg, 24 h | Cohort 3-SB-681323, 7.5 mg, 4 h | Cohort 4-SB-681323, 10 mg, 24 h
Number analyzed (Participants) | 16 | 6 | 8 | 11 | 9
pH Units | 7.358 (0.0738) | 7.363 (0.0824) | 7.358 (0.0354) | 7.353 (0.0297) | 7.373 (0.0527)

12. Primary Outcome: Vital Parameter- Mean Systolic Blood Pressure (SBP) and Diastolic Blood Pressure (DBP)
Description: Absolute values of SBP and DBP were reported.
Time Frame: For Cohort 1 and 3: "Day 1, 4 h", "Day 2, pre-dose", "Day 3, pre-dose and 24 h" and "Follow up (Day 7)"; for Cohort 2 and 4: "Day 2, pre-dose", "Day 3, pre-dose and 24 h", and "Follow up (Day 7)"
Population: All subject population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Millimeter of Mercury (mmHg)
Arm/Group | Combined Placebo | Cohort 1-SB-681323, 3 mg, 4 h | Cohort 2-SB-681323, 7.5 mg, 24 h | Cohort 3-SB-681323, 7.5 mg, 4 h | Cohort 4-SB-681323, 10 mg, 24 h
Number analyzed (Participants) | 20 | 9 | 12 | 18 | 18
Millimeter of Mercury (mmHg)
  SBP : Day 1, 4 h: number analyzed (Participants) | 9 | 9 | 0 | 18 | 0
  SBP : Day 1, 4 h | 127.9 (20.93) | 116.6 (17.33) |  | 130.4 (16.25) |
  SBP : Day 2, Pre-dose: number analyzed (Participants) | 20 | 8 | 12 | 18 | 18
  SBP : Day 2, Pre-dose | 126.4 (19.91) | 114.8 (13.72) | 130.3 (23.72) | 130.9 (24.15) | 127.1 (21.47)
  SBP : Day 3, Pre-dose: number analyzed (Participants) | 20 | 8 | 12 | 17 | 17
  SBP : Day 3, Pre-dose | 130.5 (22.65) | 119.8 (16.65) | 140.4 (35.28) | 127.9 (21.43) | 136.0 (23.57)
  SBP : Day 3, Pre-dose 24 H: number analyzed (Participants) | 20 | 8 | 12 | 17 | 17
  SBP : Day 3, Pre-dose 24 H | 138.7 (22.18) | 136.0 (23.66) | 130.3 (22.80) | 129.5 (20.23) | 128.6 (15.29)
  SBP : Follow up (Day 7) | 132.4 (19.50) | 125.5 (14.06) | 134.3 (14.10) | 132.6 (27.34) | 137.9 (18.57)
  DBP : Day 1, 4 h: number analyzed (Participants) | 9 | 9 | 0 | 18 | 0
  DBP : Day 1, 4 h | 64.6 (11.57) | 61.8 (19.44) |  | 67.6 (11.01) |
  DBP : Day 2, Pre-dose: number analyzed (Participants) | 20 | 8 | 12 | 18 | 18
  DBP : Day 2, Pre-dose | 63.9 (10.38) | 63.8 (11.57) | 58.9 (8.68) | 65.0 (12.28) | 61.7 (14.59)
  DBP : Day 3, Pre-dose: number analyzed (Participants) | 20 | 8 | 12 | 17 | 17
  DBP : Day 3, Pre-dose | 65.4 (12.04) | 63.4 (11.26) | 65.3 (13.45) | 64.6 (13.70) | 71.2 (15.42)
  DBP : Day 3, Pre-dose 24 H: number analyzed (Participants) | 20 | 8 | 12 | 17 | 17
  DBP : Day 3, Pre-dose 24 H | 69.2 (11.10) | 68.9 (10.99) | 68.9 (12.48) | 66.2 (11.09) | 74.5 (10.92)
  DBP : Follow up (Day 7): number analyzed (Participants) | 20 | 8 | 12 | 18 | 18
  DBP : Follow up (Day 7) | 66.0 (12.42) | 67.9 (12.23) | 71.0 (9.82) | 69.3 (13.31) | 74.0 (12.69)

13. Primary Outcome: Vital Parameter: Mean Heart Rate
Description: Absolute values of mean heart rate were reported.
Time Frame: as for outcome 12
Population: All subject population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Combined Placebo | Cohort 1-SB-681323, 3 mg, 4 h | Cohort 2-SB-681323, 7.5 mg, 24 h | Cohort 3-SB-681323, 7.5 mg, 4 h | Cohort 4-SB-681323, 10 mg, 24 h
Number analyzed (Participants) | 20 | 9 | 12 | 18 | 18
Beats per minute
  Heart rate: Day 1, 4 h: number analyzed (Participants) | 9 | 9 | 0 | 18 | 0
  Heart rate: Day 1, 4 h | 92.7 (12.18) | 89.7 (17.63) |  | 97.8 (15.37) |
  Heart rate: Day 2, pre-dose: number analyzed (Participants) | 20 | 8 | 11 | 18 | 18
  Heart rate: Day 2, pre-dose | 99.8 (16.92) | 93.8 (13.35) | 98.1 (27.01) | 97.1 (19.36) | 82.7 (13.52)
  Heart rate: Day 3, pre-dose: number analyzed (Participants) | 20 | 8 | 11 | 17 | 18
  Heart rate: Day 3, pre-dose | 97.0 (15.13) | 99.3 (19.90) | 88.7 (24.73) | 93.8 (12.20) | 88.3 (17.83)
  Heart rate: Day 3, 24 h: number analyzed (Participants) | 20 | 8 | 12 | 17 | 18
  Heart rate: Day 3, 24 h | 100.4 (15.20) | 99.3 (12.69) | 93.7 (16.37) | 96.4 (15.74) | 90.5 (18.49)
  Heart rate: Follow up (Day 7): number analyzed (Participants) | 20 | 8 | 12 | 18 | 18
  Heart rate: Follow up (Day 7) | 97.6 (13.42) | 93.3 (19.91) | 100.3 (18.79) | 96.8 (16.40) | 87.7 (14.09)

14. Primary Outcome: Vital Sign: Mean Percent Oxygen (O2) in Blood
Description: Absolute values of mean percent O2 in blood were reported.
Time Frame: as for outcome 12
Population: All subject population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Percent O2
Arm/Group | Combined Placebo | Cohort 1-SB-681323, 3 mg, 4 h | Cohort 2-SB-681323, 7.5 mg, 24 h | Cohort 3-SB-681323, 7.5 mg, 4 h | Cohort 4-SB-681323, 10 mg, 24 h
Number analyzed (Participants) | 20 | 9 | 12 | 18 | 18
Percent O2
  Percent O2 in blood: Day 1, 4 h: number analyzed (Participants) | 9 | 9 | 0 | 18 | 0
  Percent O2 in blood: Day 1, 4 h | 98.6 (2.30) | 97.1 (2.98) |  | 97.6 (1.65) |
  Percent O2 in blood: Day 2, pre-dose: number analyzed (Participants) | 20 | 8 | 12 | 17 | 18
  Percent O2 in blood: Day 2, pre-dose | 97.5 (2.44) | 97.3 (2.05) | 97.3 (2.87) | 96.8 (3.32) | 97.1 (3.08)
  Percent O2 in blood: Day 3, pre-dose: number analyzed (Participants) | 20 | 8 | 11 | 17 | 17
  Percent O2 in blood: Day 3, pre-dose | 97.1 (2.40) | 96.0 (4.00) | 96.9 (2.88) | 97.7 (2.49) | 96.5 (2.90)
  Percent O2 in blood: Day 3, 24 h: number analyzed (Participants) | 20 | 8 | 11 | 17 | 17
  Percent O2 in blood: Day 3, 24 h | 97.3 (2.27) | 97.9 (2.03) | 96.7 (2.41) | 97.5 (2.60) | 97.3 (2.47)
  Percent O2 in blood: Follow up (Day 7): number analyzed (Participants) | 20 | 8 | 12 | 18 | 18
  Percent O2 in blood: Follow up (Day 7) | 96.5 (2.06) | 97.3 (2.12) | 96.3 (3.11) | 97.2 (1.99) | 97.1 (1.81)

15. Primary Outcome: Vital Signs: Mean Oxygen Saturation (SaO2) Via Pulse Oximetry
Description: Assessment of SaO2 via pulse oximetry was planned for cohort 1 and 3 at Day 1 (4 h), Day 2 (pre-dose) and Day 3 (pre-dose and 24 h) and for cohort 2 and 4: Day 2 (pre-dose) and Day 3 (pre-dose and 24 h). However, the analyzable data was not collected for this parameter.
Time Frame: For Cohort 1 and 3: "Day 1, 4 h", "Day 2, pre-dose", "Day 3, pre-dose and 24 h"; for Cohort 2 and 4: "Day 2, pre-dose", and "Day 3, pre-dose and 24 h"
Population: All subject population. Data was not collected for this parameter.
Arm/Group | Combined Placebo | Cohort 1-SB-681323, 3 mg, 4 h | Cohort 2-SB-681323, 7.5 mg, 24 h | Cohort 3-SB-681323, 7.5 mg, 4 h | Cohort 4-SB-681323, 10 mg, 24 h
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

16. Primary Outcome: Vital Signs: Mean Level of Positive End Expiratory Pressure
Description: Assessment of level of positive end expiratory pressure was planned for cohort 1 and 3 at Day 1 (4 h), Day 2 (pre-dose) and Day 3 (pre-dose and 24 h) and for cohort 2 and 4: Day 2 (pre-dose) and Day 3 (pre-dose and 24 h). However, the analyzable data was not collected for this parameter.
Time Frame: as for outcome 15
Population: All subject population. Data was not collected for this parameter.
Arm/Group | Combined Placebo | Cohort 1-SB-681323, 3 mg, 4 h | Cohort 2-SB-681323, 7.5 mg, 24 h | Cohort 3-SB-681323, 7.5 mg, 4 h | Cohort 4-SB-681323, 10 mg, 24 h
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

17. Primary Outcome: Vital Signs: Mean Level of Peak and Plateau Ventilator Pressures
Description: Assessment of mean level of peak and plateau ventilator pressures was planned for cohort 1 and 3 at Day 1 (4 h), Day 2 (pre-dose) and Day 3 (pre-dose and 24 h) and for cohort 2 and 4: Day 2 (pre-dose) and Day 3 (pre-dose and 24 h). However, the analyzable data was not collected for this parameter.
Time Frame: as for outcome 15
Population: All subject population. Data was not collected for this parameter.
Arm/Group | Combined Placebo | Cohort 1-SB-681323, 3 mg, 4 h | Cohort 2-SB-681323, 7.5 mg, 24 h | Cohort 3-SB-681323, 7.5 mg, 4 h | Cohort 4-SB-681323, 10 mg, 24 h
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

18. Primary Outcome: Vital Signs: Mean Oxygen Requirement (FiO2) Via Pulse Oximetry
Description: Assessment of mean FiO2 via pulse oximetry was planned for cohort 1 and 3 at Day 1 (4 h), Day 2 (pre-dose) and Day 3 (pre-dose and 24 h) and for cohort 2 and 4: Day 2 (pre-dose) and Day 3 (pre-dose and 24 h). However, the analyzable data was not collected for this parameter.
Time Frame: as for outcome 15
Population: All subject population. Data was not collected for this parameter.
Arm/Group | Combined Placebo | Cohort 1-SB-681323, 3 mg, 4 h | Cohort 2-SB-681323, 7.5 mg, 24 h | Cohort 3-SB-681323, 7.5 mg, 4 h | Cohort 4-SB-681323, 10 mg, 24 h
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

19. Primary Outcome: Mean Electrocardiogram (ECG) Parameters Including PR, QRS, QT, and QTcB, QTcF, RR Intervals
Description: 12-lead ECGs were obtained at each timepoint during the study using an ECG machine that automatically calculated the heart rate and measures RR, PR, QRS, QT, and QTc intervals. Absolute mean values of PR, QRS, QT, and QTcB, QTcF, RR intervals were reported.
Time Frame: Day 2, pre-dose, Day 3, pre-dose, Day 3, 24 h and Follow-up (Day 7)
Population: All subject population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Milliseconds
Arm/Group | Combined Placebo | Cohort 1-SB-681323, 3 mg, 4 h | Cohort 2-SB-681323, 7.5 mg, 24 h | Cohort 3-SB-681323, 7.5 mg, 4 h | Cohort 4-SB-681323, 10 mg, 24 h
Number analyzed (Participants) | 20 | 9 | 12 | 18 | 18
Milliseconds
  PR Interval: Day 2, pre-dose: number analyzed (Participants) | 19 | 8 | 11 | 18 | 17
  PR Interval: Day 2, pre-dose | 141.4 (14.35) | 145.5 (21.21) | 141.5 (17.80) | 143.9 (30.54) | 152.9 (20.98)
  PR Interval: Day 3, pre-dose: number analyzed (Participants) | 20 | 7 | 11 | 16 | 17
  PR Interval: Day 3, pre-dose | 145.7 (20.73) | 142.0 (22.33) | 141.6 (27.43) | 148.6 (23.00) | 152.0 (25.88)
  PR Interval: Day 3, 24 h: number analyzed (Participants) | 18 | 7 | 9 | 16 | 15
  PR Interval: Day 3, 24 h | 137.0 (18.90) | 146.9 (34.15) | 142.2 (24.93) | 145.9 (21.21) | 160.7 (23.58)
  PR Interval: Follow up (Day 7): number analyzed (Participants) | 19 | 8 | 6 | 17 | 16
  PR Interval: Follow up (Day 7) | 133.9 (13.85) | 142.8 (24.33) | 142.0 (16.54) | 138.1 (26.91) | 155.1 (22.63)
  QRS Duration: Day 2, pre-dose: number analyzed (Participants) | 20 | 8 | 12 | 18 | 18
  QRS Duration: Day 2, pre-dose | 89.8 (9.26) | 86.5 (10.78) | 86.8 (12.49) | 87.2 (13.34) | 88.0 (12.63)
  QRS Duration: Day 3, pre-dose: number analyzed (Participants) | 20 | 7 | 12 | 17 | 17
  QRS Duration: Day 3, pre-dose | 90.5 (9.62) | 87.1 (8.86) | 89.5 (10.66) | 87.6 (14.56) | 86.5 (12.11)
  QRS Duration: Day 3, 24 h: number analyzed (Participants) | 18 | 7 | 10 | 16 | 16
  QRS Duration: Day 3, 24 h | 91.6 (10.48) | 85.7 (7.70) | 90.6 (8.85) | 88.3 (14.36) | 88.4 (12.29)
  QRS Duration: Follow up (Day 7): number analyzed (Participants) | 19 | 8 | 8 | 18 | 17
  QRS Duration: Follow up (Day 7) | 90.8 (9.39) | 86.0 (8.42) | 88.5 (11.35) | 85.4 (14.01) | 85.9 (10.16)
  QT Interval: Day 2, pre-dose: number analyzed (Participants) | 19 | 8 | 12 | 18 | 18
  QT Interval: Day 2, pre-dose | 338.7 (30.74) | 349.5 (29.89) | 342.0 (61.77) | 332.1 (34.00) | 365.1 (39.95)
  QT Interval: Day 3, pre-dose: number analyzed (Participants) | 20 | 7 | 12 | 17 | 16
  QT Interval: Day 3, pre-dose | 338.6 (34.99) | 352.9 (36.20) | 351.3 (56.64) | 342.5 (24.15) | 351.4 (48.51)
  QT Interval: Day 3, 24 h: number analyzed (Participants) | 18 | 7 | 10 | 16 | 16
  QT Interval: Day 3, 24 h | 328.8 (35.13) | 347.4 (28.93) | 340.2 (31.64) | 336.5 (31.22) | 358.0 (47.32)
  QT Interval: Follow up (Day 7): number analyzed (Participants) | 19 | 8 | 8 | 18 | 17
  QT Interval: Follow up (Day 7) | 346.7 (33.16) | 352.5 (16.89) | 335.0 (47.41) | 342.1 (37.14) | 369.1 (45.58)
  QTcB Interval: Day 2, pre-dose: number analyzed (Participants) | 19 | 8 | 12 | 18 | 18
  QTcB Interval: Day 2, pre-dose | 432.5 (28.82) | 427.5 (27.91) | 422.0 (28.72) | 418.6 (21.72) | 416.2 (24.28)
  QTcB Interval: Day 3, pre-dose: number analyzed (Participants) | 20 | 7 | 12 | 17 | 16
  QTcB Interval: Day 3, pre-dose | 424.4 (27.55) | 443.4 (28.77) | 414.4 (22.33) | 420.9 (26.99) | 427.4 (31.17)
  QTcB Interval: Day 3, 24 h: number analyzed (Participants) | 18 | 7 | 10 | 16 | 16
  QTcB Interval: Day 3, 24 h | 425.8 (21.83) | 425.6 (18.45) | 418.5 (22.60) | 422.5 (22.33) | 429.6 (22.05)
  QTcB Interval: Follow up (Day 7): number analyzed (Participants) | 19 | 8 | 8 | 18 | 17
  QTcB Interval: Follow up (Day 7) | 435.5 (32.08) | 439.4 (15.30) | 430.1 (43.76) | 434.7 (19.27) | 440.3 (48.93)
  QTcF Interval: Day 2, pre-dose: number analyzed (Participants) | 19 | 8 | 12 | 18 | 18
  QTcF Interval: Day 2, pre-dose | 398.3 (24.07) | 399.4 (22.88) | 392.6 (36.62) | 387.1 (22.19) | 397.9 (24.09)
  QTcF Interval: Day 3, pre-dose: number analyzed (Participants) | 20 | 7 | 12 | 17 | 16
  QTcF Interval: Day 3, pre-dose | 393.3 (27.85) | 410.5 (26.01) | 391.5 (30.90) | 392.7 (21.41) | 400.0 (35.34)
  QTcF Interval: Day 3, 24 h: number analyzed (Participants) | 18 | 7 | 10 | 16 | 16
  QTcF Interval: Day 3, 24 h | 390.4 (24.77) | 397.4 (14.85) | 390.3 (22.25) | 391.4 (22.27) | 403.7 (26.80)
  QTcF Interval: Follow up (Day 7): number analyzed (Participants) | 19 | 8 | 8 | 18 | 17
  QTcF Interval: Follow up (Day 7) | 403.4 (29.35) | 408.1 (11.78) | 395.5 (43.63) | 401.0 (23.91) | 414.9 (45.44)
  RR Interval: Day 2, pre-dose: number analyzed (Participants) | 19 | 8 | 12 | 18 | 18
  RR Interval: Day 2, pre-dose | 622.0 (117.16) | 677.5 (133.48) | 667.7 (219.26) | 635.5 (119.09) | 780.8 (178.59)
  RR Interval: Day 3, pre-dose: number analyzed (Participants) | 20 | 7 | 12 | 17 | 16
  RR Interval: Day 3, pre-dose | 640.1 (103.46) | 641.4 (137.62) | 727.9 (210.54) | 670.2 (115.37) | 679.5 (140.86)
  RR Interval: Day 3, 24 h: number analyzed (Participants) | 18 | 7 | 10 | 16 | 16
  RR Interval: Day 3, 24 h | 598.7 (99.54) | 675.1 (137.03) | 665.8 (114.27) | 639.0 (106.37) | 703.1 (171.59)
  RR Interval: Follow up (Day 7): number analyzed (Participants) | 19 | 8 | 8 | 18 | 17
  RR Interval: Follow up (Day 7) | 639.0 (103.45) | 646.8 (74.52) | 608.3 (98.05) | 622.3 (105.38) | 709.0 (112.18)

20. Primary Outcome: Number of Participants With Any Adverse Events (AE) and Serious Adverse Events (SAE)
Description: AE was defined as any untoward medical occurrence in a participant temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. SAE include AEs those result in death, a life-threatening AE, inpatient hospitalization or prolongation of existing hospitalization, a persistent or significant incapacity or substantial disruption of the ability to conduct normal functions, or a congenital anomaly/birth defect. Important medical events that may not result in death, be life-threatening, or require hospitalization may be considered serious when, based upon appropriate medical judgment, they may jeopardize the participant and may require medical or surgical intervention to prevent one of the outcomes listed in this definition.
Time Frame: Up to Follow-up (Day 7)
Population: All subject population.
Measure: Count of Participants; unit: Participants
Arm/Group | Combined Placebo | Cohort 1-SB-681323, 3 mg, 4 h | Cohort 2-SB-681323, 7.5 mg, 24 h | Cohort 3-SB-681323, 7.5 mg, 4 h | Cohort 4-SB-681323, 10 mg, 24 h
Number analyzed (Participants) | 20 | 9 | 12 | 18 | 18
Participants
  Any AEs | 18 | 7 | 10 | 16 | 14
  Any SAEs | 1 | 1 | 1 | 4 | 0

21. Secondary Outcome: Mean Serum Interleukin-6 Levels
Description: Serum samples were collected at 6, 12, 18, 24, 48, 72 and 96 h since first dose on Day 1. Mean absolute values of Serum interleukin-6 levels at these specified time oints were reported.
Time Frame: 6, 12, 18, 24, 48, 72 and 96 h since first dose on Day 1
Population: Pharmacodynamic (PD) Population was defined as patients in the 'All Subjects' population for whom a pharmacodynamic sample was obtained and analysed (Flow Cytometry data were excluded from the definition of pharmacodynamic sample). Only those participants available at the specified time points were analyzed.
Measure: Geometric Mean (95% Confidence Interval); unit: Picogram per milliliter (pg/mL)
Arm/Group | Combined Placebo | Cohort 1-SB-681323, 3 mg, 4 h | Cohort 2-SB-681323, 7.5 mg, 24 h | Cohort 3-SB-681323, 7.5 mg, 4 h | Cohort 4-SB-681323, 10 mg, 24 h
Number analyzed (Participants) | 20 | 8 | 10 | 16 | 18
Picogram per milliliter (pg/mL)
  Time Since 1st Dose, 6 h: number analyzed (Participants) | 18 | 6 | 10 | 16 | 18
  Time Since 1st Dose, 6 h | 509.44 [404.31 to 641.92] | 286.17 [193.56 to 423.09] | 391.09 [285.50 to 535.73] | 309.57 [241.39 to 397.00] | 395.09 [311.51 to 501.11]
  Time Since 1st Dose, 12 h: number analyzed (Participants) | 19 | 7 | 10 | 15 | 17
  Time Since 1st Dose, 12 h | 516.49 [386.08 to 690.93] | 315.89 [195.60 to 510.16] | 362.03 [242.29 to 540.95] | 348.23 [252.52 to 480.21] | 310.98 [229.12 to 422.08]
  Time Since 1st Dose, 18 h: number analyzed (Participants) | 19 | 7 | 10 | 14 | 18
  Time Since 1st Dose, 18 h | 476.94 [342.58 to 663.98] | 247.22 [143.35 to 426.37] | 275.7 [174.63 to 435.27] | 292.24 [202.25 to 422.28] | 238.7 [167.94 to 339.28]
  Time Since 1st Dose, 24 h: number analyzed (Participants) | 19 | 7 | 10 | 15 | 17
  Time Since 1st Dose, 24 h | 556.06 [396.84 to 779.16] | 231.1 [132.58 to 402.84] | 228.1 [143.19 to 363.33] | 310.47 [214.22 to 449.97] | 162.82 [111.89 to 236.94]
  Time Since 1st Dose, 48 h: number analyzed (Participants) | 19 | 7 | 9 | 15 | 16
  Time Since 1st Dose, 48 h | 324.35 [227.93 to 461.57] | 167.69 [93.79 to 299.85] | 290.59 [175.53 to 481.08] | 235.13 [158.44 to 348.94] | 119.98 [75.81 to 189.87]
  Time Since 1st Dose, 72 h: number analyzed (Participants) | 17 | 7 | 9 | 15 | 13
  Time Since 1st Dose, 72 h | 250.21 [162.45 to 385.39] | 165.46 [82.36 to 332.41] | 184.93 [100.25 to 341.14] | 182.54 [113.18 to 294.40] | 106.32 [62.32 to 181.39]
  Time Since 1st Dose, 96 h: number analyzed (Participants) | 17 | 7 | 7 | 14 | 13
  Time Since 1st Dose, 96 h | 183.79 [113.50 to 297.61] | 166.87 [77.25 to 360.46] | 286.79 [139.88 to 587.97] | 210.87 [123.37 to 360.41] | 106.32 [62.32 to 181.39]
Statistical Analysis 1: Comparison: Combined Placebo vs Cohort 1-SB-681323, 3 mg, 4 h; Comparison at 6 h post first dose; Test type: Superiority or Other; Ratio (Treatment/Placebo) = 0.562, 95% CI 2-sided [0.357 to 0.885], Standard Error of Mean 0.228
Statistical Analysis 2: Comparison: Combined Placebo vs Cohort 1-SB-681323, 3 mg, 4 h; Comparison at 12 h post first dose; Test type: Superiority or Other; Ratio (Treatment/Placebo) = 0.612, 95% CI 2-sided [0.349 to 1.072], Standard Error of Mean 0.281
Statistical Analysis 3: Comparison: Combined Placebo vs Cohort 1-SB-681323, 3 mg, 4 h; Comparison at 18 h post first dose; Test type: Superiority or Other; Ratio (Treatment/Placebo) = 0.518, 95% CI 2-sided [0.274 to 0.981], Standard Error of Mean 0.319
Statistical Analysis 4: Comparison: Combined Placebo vs Cohort 1-SB-681323, 3 mg, 4 h; Comparison at 24 h post first dose; Test type: Superiority or Other; Ratio (Treatment/Placebo) = 0.416, 95% CI 2-sided [0.217 to 0.796], Standard Error of Mean 0.326
Statistical Analysis 5: Comparison: Combined Placebo vs Cohort 1-SB-681323, 3 mg, 4 h; Comparison at 48 h post first dose; Test type: Superiority or Other; Ratio (Treatment/Placebo) = 0.517, 95% CI 2-sided [0.262 to 1.021], Standard Error of Mean 0.340
Statistical Analysis 6: Comparison: Combined Placebo vs Cohort 1-SB-681323, 3 mg, 4 h; Comparison at 72 h post first dose; Test type: Superiority or Other; Ratio (Treatment/Placebo) = 0.661, 95% CI 2-sided [0.291 to 1.503], Standard Error of Mean 0.410
Statistical Analysis 7: Comparison: Combined Placebo vs Cohort 1-SB-681323, 3 mg, 4 h; Comparison at 96 h post first dose; Test type: Superiority or Other; Ratio (Treatment/Placebo) = 0.908, 95% CI 2-sided [0.366 to 2.254], Standard Error of Mean 0.454
Statistical Analysis 8: Comparison: Combined Placebo vs Cohort 2-SB-681323, 7.5 mg, 24 h; Comparison at 6 h post first dose; Test type: Superiority or Other; Ratio (Treatment/Placebo) = 0.768, 95% CI 2-sided [0.520 to 1.134], Standard Error of Mean 0.195
Statistical Analysis 9: Comparison: Combined Placebo vs Cohort 2-SB-681323, 7.5 mg, 24 h; Comparison at 12 h post first dose; Test type: Superiority or Other; Ratio (Treatment/Placebo) = 0.701, 95% CI 2-sided [0.427 to 1.150], Standard Error of Mean 0.248
Statistical Analysis 10: Comparison: Combined Placebo vs Cohort 2-SB-681323, 7.5 mg, 24 h; Comparison at 18 h post first dose; Test type: Superiority or Other; Ratio (Treatment/Placebo) = 0.578, 95% CI 2-sided [0.329 to 1.015], Standard Error of Mean 0.282
Statistical Analysis 11: Comparison: Combined Placebo vs Cohort 2-SB-681323, 7.5 mg, 24 h; Comparison at 24 h post first dose; Test type: Superiority or Other; Ratio (Treatment/Placebo) = 0.410, 95% CI 2-sided [0.231 to 0.728], Standard Error of Mean 0.287
Statistical Analysis 12: Comparison: Combined Placebo vs Cohort 2-SB-681323, 7.5 mg, 24 h; Comparison at 48 h post first dose; Test type: Superiority or Other; Ratio (Treatment/Placebo) = 0.896, 95% CI 2-sided [0.484 to 1.657], Standard Error of Mean 0.308
Statistical Analysis 13: Comparison: Combined Placebo vs Cohort 2-SB-681323, 7.5 mg, 24 h; Comparison at 72 h post first dose; Test type: Superiority or Other; Ratio (Treatment/Placebo) = 0.739, 95% CI 2-sided [0.350 to 1.563], Standard Error of Mean 0.374
Statistical Analysis 14: Comparison: Combined Placebo vs Cohort 2-SB-681323, 7.5 mg, 24 h; Comparison at 96 h post first dose; Test type: Superiority or Other; Ratio (Treatment/Placebo) = 1.560, 95% CI 2-sided [0.659 to 3.697], Standard Error of Mean 0.431
Statistical Analysis 15: Comparison: Combined Placebo vs Cohort 3-SB-681323, 7.5 mg, 4 h; Comparison at 6 h post first dose; Test type: Superiority or Other; Ratio (Treatment/Placebo) = 0.608, 95% CI 2-sided [0.433 to 0.853], Standard Error of Mean 0.170
Statistical Analysis 16: Comparison: Combined Placebo vs Cohort 3-SB-681323, 7.5 mg, 4 h; Comparison at 12 h post first dose; Test type: Superiority or Other; Ratio (Treatment/Placebo) = 0.674, 95% CI 2-sided [0.437 to 1.039], Standard Error of Mean 0.217
Statistical Analysis 17: Comparison: Combined Placebo vs Cohort 3-SB-681323, 7.5 mg, 4 h; Comparison at 18 h post first dose; Test type: Superiority or Other; Ratio (Treatment/Placebo) = 0.613, 95% CI 2-sided [0.374 to 1.004], Standard Error of Mean 0.247
Statistical Analysis 18: Comparison: Combined Placebo vs Cohort 3-SB-681323, 7.5 mg, 4 h; Comparison at 24 h post first dose; Test type: Superiority or Other; Ratio (Treatment/Placebo) = 0.558, 95% CI 2-sided [0.338 to 0.921], Standard Error of Mean 0.251
Statistical Analysis 19: Comparison: Combined Placebo vs Cohort 3-SB-681323, 7.5 mg, 4 h; Comparison at 48 h post first dose; Test type: Superiority or Other; Ratio (Treatment/Placebo) = 0.725, 95% CI 2-sided [0.427 to 1.230], Standard Error of Mean 0.264
Statistical Analysis 20: Comparison: Combined Placebo vs Cohort 3-SB-681323, 7.5 mg, 4 h; Comparison at 72 h post first dose; Test type: Superiority or Other; Ratio (Treatment/Placebo) = 0.730, 95% CI 2-sided [0.384 to 1.386], Standard Error of Mean 0.321
Statistical Analysis 21: Comparison: Combined Placebo vs Cohort 3-SB-681323, 7.5 mg, 4 h; Comparison at 96 h post first dose; Test type: Superiority or Other; Ratio (Treatment/Placebo) = 1.147, 95% CI 2-sided [0.559 to 2.353], Standard Error of Mean 0.359
Statistical Analysis 22: Comparison: Combined Placebo vs Cohort 4-SB-681323, 10 mg, 24 h; Comparison at 6 h post first dose; Test type: Superiority or Other; Ratio (Treatment/Placebo) = 0.776, 95% CI 2-sided [0.556 to 1.082], Standard Error of Mean 0.167
Statistical Analysis 23: Comparison: Combined Placebo vs Cohort 4-SB-681323, 10 mg, 24 h; Comparison at 12 h post first dose; Test type: Superiority or Other; Ratio (Treatment/Placebo) = 0.602, 95% CI 2-sided [0.394 to 0.919], Standard Error of Mean 0.212
Statistical Analysis 24: Comparison: Combined Placebo vs Cohort 4-SB-681323, 10 mg, 24 h; Comparison at 18 h post first dose; Test type: Superiority or Other; Ratio (Treatment/Placebo) = 0.623, 95% CI 2-sided [0.386 to 1.007], Standard Error of Mean 0.240
Statistical Analysis 25: Comparison: Combined Placebo vs Cohort 4-SB-681323, 10 mg, 24 h; Comparison at 24 h post first dose; Test type: Superiority or Other; Ratio (Treatment/Placebo) = 0.429, 95% CI 2-sided [0.263 to 0.700], Standard Error of Mean 0.245
Statistical Analysis 26: Comparison: Combined Placebo vs Cohort 4-SB-681323, 10 mg, 24 h; Comparison at 48 h post first dose; Test type: Superiority or Other; Ratio (Treatment/Placebo) = 0.502, 95% CI 2-sided [0.299 to 0.842], Standard Error of Mean 0.259
Statistical Analysis 27: Comparison: Combined Placebo vs Cohort 4-SB-681323, 10 mg, 24 h; Comparison at 72 h post first dose; Test type: Superiority or Other; Ratio (Treatment/Placebo) = 0.479, 95% CI 2-sided [0.255 to 0.903], Standard Error of Mean 0.317
Statistical Analysis 28: Comparison: Combined Placebo vs Cohort 4-SB-681323, 10 mg, 24 h; Comparison at 96 h post first dose; Test type: Superiority or Other; Ratio (Treatment/Placebo) = 0.579, 95% CI 2-sided [0.281 to 1.192], Standard Error of Mean 0.361

22. Secondary Outcome: Mean Serum CXCL8 (Interleuin-8) Levels
Description: Serum samples were collected at 6, 12, 18, 24, 48, 72 and 96 h since first dose on Day 1. Mean absolute values of Serum CXCL8 (Interleuin-8) levels at these specified time points were reported.
Time Frame: 6, 12, 18, 24, 48, 72 and 96 h since first dose on Day 1
Population: PD Population. Only those participants available at the specified time points were analyzed.
Measure: Geometric Mean (95% Confidence Interval); unit: pg/ml
Arm/Group | Combined Placebo | Cohort 1-SB-681323, 3 mg, 4 h | Cohort 2-SB-681323, 7.5 mg, 24 h | Cohort 3-SB-681323, 7.5 mg, 4 h | Cohort 4-SB-681323, 10 mg, 24 h
Number analyzed (Participants) | 20 | 8 | 10 | 16 | 18
pg/ml
  Time Since 1st Dose, 6 h: number analyzed (Participants) | 17 | 7 | 10 | 16 | 18
  Time Since 1st Dose, 6 h | 37.66 [29.86 to 47.50] | 18.22 [12.53 to 26.50] | 27.34 [19.88 to 37.60] | 21.06 [16.53 to 26.84] | 21.85 [17.38 to 27.46]
  Time Since 1st Dose, 12 h: number analyzed (Participants) | 19 | 7 | 10 | 15 | 17
  Time Since 1st Dose, 12 h | 26.53 [19.86 to 35.44] | 18.58 [11.42 to 30.21] | 21.00 [13.88 to 31.77] | 22.01 [16.00 to 30.29] | 17.42 [12.89 to 23.53]
  Time Since 1st Dose, 18 h: number analyzed (Participants) | 19 | 7 | 10 | 13 | 18
  Time Since 1st Dose, 18 h | 21.37 [15.61 to 29.26] | 14.55 [8.59 to 24.67] | 15.49 [9.88 to 24.28] | 21.10 [14.76 to 30.16] | 15.96 [11.57 to 22.04]
  Time Since 1st Dose, 24 h: number analyzed (Participants) | 19 | 7 | 10 | 15 | 18
  Time Since 1st Dose, 24 h | 24.05 [17.63 to 32.81] | 16.19 [9.61 to 27.28] | 15.75 [10.10 to 24.54] | 22.23 [15.79 to 31.29] | 15.79 [11.48 to 21.72]
  Time Since 1st Dose, 48 h: number analyzed (Participants) | 19 | 7 | 9 | 15 | 17
  Time Since 1st Dose, 48 h | 17.65 [12.30 to 25.33] | 16.24 [8.85 to 29.80] | 19.62 [11.55 to 33.32] | 21.70 [14.54 to 32.41] | 13.40 [9.19 to 19.53]
  Time Since 1st Dose, 72 h: number analyzed (Participants) | 17 | 7 | 9 | 14 | 16
  Time Since 1st Dose, 72 h | 15.99 [10.80 to 23.66] | 15.09 [7.91 to 28.75] | 17.19 [9.76 to 30.26] | 20.61 [13.36 to 31.77] | 15.47 [10.30 to 23.23]
  Time Since 1st Dose, 96 h: number analyzed (Participants) | 17 | 7 | 7 | 13 | 13
  Time Since 1st Dose, 96 h | 19.14 [13.65 to 26.84] | 17.33 [9.99 to 30.06] | 26.32 [15.58 to 44.47] | 33.54 [22.92 to 49.08] | 14.24 [9.81 to 20.65]
Statistical Analysis 1: Comparison: Combined Placebo vs Cohort 1-SB-681323, 3 mg, 4 h; Comparison at 6 h post first dose; Test type: Superiority or Other; Ratio (Treatment/Placebo) = 0.484, 95% CI 2-sided [0.312 to 0.750], Standard Error of Mean 0.219
Statistical Analysis 2: Comparison: Combined Placebo vs Cohort 1-SB-681323, 3 mg, 4 h; Comparison at 12 h post first dose; Test type: Superiority or Other; Ratio (Treatment/Placebo) = 0.700, 95.000% CI 2-sided [0.399 to 1.229], Standard Error of Mean 0.282
Statistical Analysis 3: Comparison: Combined Placebo vs Cohort 1-SB-681323, 3 mg, 4 h; Comparison at 18 h post first dose; Test type: Superiority or Other; Ratio (Treatment/Placebo) = 0.681, 95.000% CI 2-sided [0.370 to 1.254], Standard Error of Mean 0.305
Statistical Analysis 4: Comparison: Combined Placebo vs Cohort 1-SB-681323, 3 mg, 4 h; Comparison at 24 h post first dose; Test type: Superiority or Other; Ratio (Treatment/Placebo) = 0.673, 95.000% CI 2-sided [0.368 to 1.231], Standard Error of Mean 0.302
Statistical Analysis 5: Comparison: Combined Placebo vs Cohort 1-SB-681323, 3 mg, 4 h; Comparison at 48 h post first dose; Test type: Superiority or Other; Ratio (Treatment/Placebo) = 0.920, 95.000% CI 2-sided [0.456 to 1.857], Standard Error of Mean 0.351
Statistical Analysis 6: Comparison: Combined Placebo vs Cohort 1-SB-681323, 3 mg, 4 h; Comparison at 72 h post first dose; Test type: Superiority or Other; Ratio (Treatment/Placebo) = 0.944, 95.000% CI 2-sided [0.445 to 2.002], Standard Error of Mean 0.376
Statistical Analysis 7: Comparison: Combined Placebo vs Cohort 1-SB-681323, 3 mg, 4 h; Comparison at 96 h post first dose; Test type: Superiority or Other; Ratio (Treatment/Placebo) = 0.905, 95.000% CI 2-sided [0.476 to 1.723], Standard Error of Mean 0.321
Statistical Analysis 8: Comparison: Combined Placebo vs Cohort 2-SB-681323, 7.5 mg, 24 h; Comparison at 6 h post first dose; Test type: Superiority or Other; Ratio (Treatment/Placebo) = 0.726, 95.000% CI 2-sided [0.488 to 1.080], Standard Error of Mean 0.199
Statistical Analysis 9: Comparison: Combined Placebo vs Cohort 2-SB-681323, 7.5 mg, 24 h; Comparison at 12 h post first dose; Test type: Superiority or Other; Ratio (Treatment/Placebo) = 0.791, 95.000% CI 2-sided [0.476 to 1.317], Standard Error of Mean 0.255
Statistical Analysis 10: Comparison: Combined Placebo vs Cohort 2-SB-681323, 7.5 mg, 24 h; Comparison at 18 h post first dose; Test type: Superiority or Other; Ratio (Treatment/Placebo) = 0.725, 95.000% CI 2-sided [0.417 to 1.260], Standard Error of Mean 0.277
Statistical Analysis 11: Comparison: Combined Placebo vs Cohort 2-SB-681323, 7.5 mg, 24 h; Comparison at 24 h post first dose; Test type: Superiority or Other; Ratio (Treatment/Placebo) = 0.655, 95.000% CI 2-sided [0.379 to 1.130], Standard Error of Mean 0.273
Statistical Analysis 12: Comparison: Combined Placebo vs Cohort 2-SB-681323, 7.5 mg, 24 h; Comparison at 48 h post first dose; Test type: Superiority or Other; Ratio (Treatment/Placebo) = 1.111, 95.000% CI 2-sided [0.583 to 2.120], Standard Error of Mean 0.323
Statistical Analysis 13: Comparison: Combined Placebo vs Cohort 2-SB-681323, 7.5 mg, 24 h; Comparison at 72 h post first dose; Test type: Superiority or Other; Ratio (Treatment/Placebo) = 1.075, 95.000% CI 2-sided [0.539 to 2.146], Standard Error of Mean 0.346
Statistical Analysis 14: Comparison: Combined Placebo vs Cohort 2-SB-681323, 7.5 mg, 24 h; Comparison at 96 h post first dose; Test type: Superiority or Other; Ratio (Treatment/Placebo) = 1.375, 95.000% CI 2-sided [0.735 to 2.574], Standard Error of Mean 0.313
Statistical Analysis 15: Comparison: Combined Placebo vs Cohort 3-SB-681323, 7.5 mg, 4 h; Comparison at 6 h post first dose; Test type: Superiority or Other; Ratio (Treatment/Placebo) = 0.559, 95.000% CI 2-sided [0.400 to 0.783], Standard Error of Mean 0.168
Statistical Analysis 16: Comparison: Combined Placebo vs Cohort 3-SB-681323, 7.5 mg, 4 h; Comparison at 12 h post first dose; Test type: Superiority or Other; Ratio (Treatment/Placebo) = 0.830, 95.000% CI 2-sided [0.539 to 1.277], Standard Error of Mean 0.216
Statistical Analysis 17: Comparison: Combined Placebo vs Cohort 3-SB-681323, 7.5 mg, 4 h; Comparison at 18 h post first dose; Test type: Superiority or Other; Ratio (Treatment/Placebo) = 0.987, 95.00% CI 2-sided [0.613 to 1.589], Standard Error of Mean 0.238
Statistical Analysis 18: Comparison: Combined Placebo vs Cohort 3-SB-681323, 7.5 mg, 4 h; Comparison at 24 h post first dose; Test type: Superiority or Other; Ratio (Treatment/Placebo) = 0.924, 95.00% CI 2-sided [0.582 to 1.467], Standard Error of Mean 0.231
Statistical Analysis 19: Comparison: Combined Placebo vs Cohort 3-SB-681323, 7.5 mg, 4 h; Comparison at 48 h post first dose; Test type: Superiority or Other; Ratio (Treatment/Placebo) = 1.230, 95.00% CI 2-sided [0.716 to 2.110], Standard Error of Mean 0.270
Statistical Analysis 20: Comparison: Combined Placebo vs Cohort 3-SB-681323, 7.5 mg, 4 h; Comparison at 72 h post first dose; Test type: Superiority or Other; Ratio (Treatment/Placebo) = 1.289, 95.00% CI 2-sided [0.719 to 2.312], Standard Error of Mean 0.292
Statistical Analysis 21: Comparison: Combined Placebo vs Cohort 3-SB-681323, 7.5 mg, 4 h; Comparison at 96 h post first dose; Test type: Superiority or Other; Ratio (Treatment/Placebo) = 1.752, 95.00% CI 2-sided [1.053 to 2.916], Standard Error of Mean 0.254
Statistical Analysis 22: Comparison: Combined Placebo vs Cohort 4-SB-681323, 10 mg, 24 h; Comparison at 6 h post first dose; Test type: Superiority or Other; Ratio (Treatment/Placebo) = 0.580, 95.00% CI 2-sided [0.419 to 0.803], Standard Error of Mean 0.163
Statistical Analysis 23: Comparison: Combined Placebo vs Cohort 4-SB-681323, 10 mg, 24 h; Comparison at 12 h post first dose; Test type: Superiority or Other; Ratio (Treatment/Placebo) = 0.657, 95.00% CI 2-sided [0.433 to 0.996], Standard Error of Mean 0.209
Statistical Analysis 24: Comparison: Combined Placebo vs Cohort 4-SB-681323, 10 mg, 24 h; Comparison at 18 h post first dose; Test type: Superiority or Other; Ratio (Treatment/Placebo) = 0.747, 95.00% CI 2-sided [0.477 to 1.171], Standard Error of Mean 0.225
Statistical Analysis 25: Comparison: Combined Placebo vs Cohort 4-SB-681323, 10 mg, 24 h; Comparison at 24 h post first dose; Test type: Superiority or Other; Ratio (Treatment/Placebo) = 0.657, 95.00% CI 2-sided [0.421 to 1.024], Standard Error of Mean 0.222
Statistical Analysis 26: Comparison: Combined Placebo vs Cohort 4-SB-681323, 10 mg, 24 h; Comparison at 48 h post first dose; Test type: Superiority or Other; Ratio (Treatment/Placebo) = 0.759, 95.00% CI 2-sided [0.451 to 1.279], Standard Error of Mean 0.261
Statistical Analysis 27: Comparison: Combined Placebo vs Cohort 4-SB-681323, 10 mg, 24 h; Comparison at 72 h post first dose; Test type: Superiority or Other; Ratio (Treatment/Placebo) = 0.968, 95.00% CI 2-sided [0.550 to 1.701], Standard Error of Mean 0.282
Statistical Analysis 28: Comparison: Combined Placebo vs Cohort 4-SB-681323, 10 mg, 24 h; Comparison at 96 h post first dose; Test type: Superiority or Other; Ratio (Treatment/Placebo) = 0.744, 95.00% CI 2-sided [0.450 to 1.229], Standard Error of Mean 0.251

23. Secondary Outcome: Mean Serum C-Reactive Protein (CRP) Levels
Description: Serum samples were collected at 6, 12, 18, 24, 48, 72 and 96 h since first dose on Day 1. Mean absolute values of serum CRP levels at these specified time points were reported.
Time Frame: 6, 12, 18, 24, 48, 72 and 96 h since first dose on Day 1
Population: PD Population. Only those participants available at the specified time points were analyzed.
Measure: Geometric Mean (95% Confidence Interval); unit: mg/L
Arm/Group | Combined Placebo | Cohort 1-SB-681323, 3 mg, 4 h | Cohort 2-SB-681323, 7.5 mg, 24 h | Cohort 3-SB-681323, 7.5 mg, 4 h | Cohort 4-SB-681323, 10 mg, 24 h
Number analyzed (Participants) | 20 | 8 | 10 | 16 | 18
mg/L
  Time Since 1st Dose, 6 h: number analyzed (Participants) | 18 | 7 | 10 | 16 | 18
  Time Since 1st Dose, 6 h | 123.62 [108.90 to 140.33] | 95.60 [77.82 to 117.45] | 117.68 [99.05 to 139.82] | 117.42 [102.48 to 134.55] | 110.88 [97.49 to 126.10]
  Time Since 1st Dose, 12 h: number analyzed (Participants) | 19 | 7 | 10 | 16 | 17
  Time Since 1st Dose, 12 h | 138.02 [117.47 to 162.17] | 109.74 [84.28 to 142.88] | 133.17 [106.76 to 166.11] | 136.01 [114.22 to 161.96] | 122.42 [103.71 to 144.52]
  Time Since 1st Dose, 18 h: number analyzed (Participants) | 19 | 7 | 10 | 15 | 18
  Time Since 1st Dose, 18 h | 144.10 [118.34 to 175.45] | 112.06 [81.18 to 154.69] | 142.96 [109.14 to 187.25] | 153.76 [123.93 to 190.78] | 121.97 [99.71 to 149.20]
  Time Since 1st Dose, 24 h: number analyzed (Participants) | 19 | 7 | 10 | 16 | 18
  Time Since 1st Dose, 24 h | 153.88 [125.86 to 188.14] | 97.42 [70.10 to 135.38] | 140.47 [106.64 to 185.04] | 141.84 [114.09 to 176.33] | 125.02 [101.78 to 153.57]
  Time Since 1st Dose, 48 h: number analyzed (Participants) | 19 | 7 | 8 | 15 | 17
  Time Since 1st Dose, 48 h | 159.36 [122.11 to 207.97] | 105.45 [68.22 to 162.98] | 105.17 [71.94 to 153.77] | 138.05 [103.11 to 184.84] | 92.50 [70.13 to 122.02]
  Time Since 1st Dose, 72 h: number analyzed (Participants) | 17 | 7 | 9 | 15 | 16
  Time Since 1st Dose, 72 h | 179.03 [138.38 to 231.62] | 83.21 [55.09 to 125.67] | 123.58 [86.64 to 176.27] | 116.27 [88.06 to 153.52] | 78.55 [60.09 to 102.69]
  Time Since 1st Dose, 96 h: number analyzed (Participants) | 17 | 7 | 7 | 14 | 12
  Time Since 1st Dose, 96 h | 171.67 [126.16 to 233.62] | 90.20 [55.50 to 146.58] | 124.33 [80.24 to 192.64] | 123.97 [88.87 to 172.95] | 77.40 [55.46 to 108.01]
Statistical Analysis 1: Comparison: Combined Placebo vs Cohort 1-SB-681323, 3 mg, 4 h; Comparison at 6 h post first dose; Test type: Superiority or Other; Ratio (Treatment/Placebo) = 0.773, 95.00% CI 2-sided [0.607 to 0.985], Standard Error of Mean 0.121
Statistical Analysis 2: Comparison: Combined Placebo vs Cohort 1-SB-681323, 3 mg, 4 h; Comparison at 12 h post first dose; Test type: Superiority or Other; Ratio (Treatment/Placebo) = 0.795, 95.00% CI 2-sided [0.583 to 1.084], Standard Error of Mean 0.155
Statistical Analysis 3: Comparison: Combined Placebo vs Cohort 1-SB-681323, 3 mg, 4 h; Comparison at 18 h post first dose; Test type: Superiority or Other; Ratio (Treatment/Placebo) = 0.778, 95.00% CI 2-sided [0.533 to 1.135], Standard Error of Mean 0.189
Statistical Analysis 4: Comparison: Combined Placebo vs Cohort 1-SB-681323, 3 mg, 4 h; Comparison at 24 h post first dose; Test type: Superiority or Other; Ratio (Treatment/Placebo) = 0.633, 95.00% CI 2-sided [0.430 to 0.931], Standard Error of Mean 0.193
Statistical Analysis 5: Comparison: Combined Placebo vs Cohort 1-SB-681323, 3 mg, 4 h; Comparison at 48 h post first dose; Test type: Superiority or Other; Ratio (Treatment/Placebo) = 0.662, 95.00% CI 2-sided [0.397 to 1.103], Standard Error of Mean 0.255
Statistical Analysis 6: Comparison: Combined Placebo vs Cohort 1-SB-681323, 3 mg, 4 h; Comparison at 72 h post first dose; Test type: Superiority or Other; Ratio (Treatment/Placebo) = 0.465, 95.00% CI 2-sided [0.286 to 0.756], Standard Error of Mean 0.243
Statistical Analysis 7: Comparison: Combined Placebo vs Cohort 1-SB-681323, 3 mg, 4 h; Comparison at 96 h post first dose; Test type: Superiority or Other; Ratio (Treatment/Placebo) = 0.525, 95.00% CI 2-sided [0.295 to 0.935], Standard Error of Mean 0.287
Statistical Analysis 8: Comparison: Combined Placebo vs Cohort 2-SB-681323, 7.5 mg, 24 h; Comparison at 6 h post first dose; Test type: Superiority or Other; Ratio (Treatment/Placebo) = 0.952, 95.00% CI 2-sided [0.768 to 1.180], Standard Error of Mean 0.107
Statistical Analysis 9: Comparison: Combined Placebo vs Cohort 2-SB-681323, 7.5 mg, 24 h; Comparison at 12 h post first dose; Test type: Superiority or Other; Ratio (Treatment/Placebo) = 0.965, 95.00% CI 2-sided [0.733 to 1.269], Standard Error of Mean 0.137
Statistical Analysis 10: Comparison: Combined Placebo vs Cohort 2-SB-681323, 7.5 mg, 24 h; Comparison at 18 h post first dose; Test type: Superiority or Other; Ratio (Treatment/Placebo) = 0.992, 95.00% CI 2-sided [0.710 to 1.387], Standard Error of Mean 0.168
Statistical Analysis 11: Comparison: Combined Placebo vs Cohort 2-SB-681323, 7.5 mg, 24 h; Comparison at 24 h post first dose; Test type: Superiority or Other; Ratio (Treatment/Placebo) = 0.913, 95.00% CI 2-sided [0.649 to 1.285], Standard Error of Mean 0.171
Statistical Analysis 12: Comparison: Combined Placebo vs Cohort 2-SB-681323, 7.5 mg, 24 h; Comparison at 48 h post first dose; Test type: Superiority or Other; Ratio (Treatment/Placebo) = 0.660, 95.00% CI 2-sided [0.415 to 1.051], Standard Error of Mean 0.233
Statistical Analysis 13: Comparison: Combined Placebo vs Cohort 2-SB-681323, 7.5 mg, 24 h; Comparison at 72 h post first dose; Test type: Superiority or Other; Ratio (Treatment/Placebo) = 0.690, 95.00% CI 2-sided [0.445 to 1.072], Standard Error of Mean 0.220
Statistical Analysis 14: Comparison: Combined Placebo vs Cohort 2-SB-681323, 7.5 mg, 24 h; Comparison at 96 h post first dose; Test type: Superiority or Other; Ratio (Treatment/Placebo) = 0.724, 95.00% CI 2-sided [0.423 to 1.239], Standard Error of Mean 0.268
Statistical Analysis 15: Comparison: Combined Placebo vs Cohort 3-SB-681323, 7.5 mg, 4 h; Comparison at 6 h post first dose; Test type: Superiority or Other; Ratio (Treatment/Placebo) = 0.950, 95.00% CI 2-sided [0.789 to 1.144], Standard Error of Mean 0.093
Statistical Analysis 16: Comparison: Combined Placebo vs Cohort 3-SB-681323, 7.5 mg, 4 h; Comparison at 12 h post first dose; Test type: Superiority or Other; Ratio (Treatment/Placebo) = 0.985, 95.00% CI 2-sided [0.777 to 1.249], Standard Error of Mean 0.119
Statistical Analysis 17: Comparison: Combined Placebo vs Cohort 3-SB-681323, 7.5 mg, 4 h; Comparison at 18 h post first dose; Test type: Superiority or Other; Ratio (Treatment/Placebo) = 1.067, 95.00% CI 2-sided [0.797 to 1.428], Standard Error of Mean 0.146
Statistical Analysis 18: Comparison: Combined Placebo vs Cohort 3-SB-681323, 7.5 mg, 4 h; Comparison at 24 h post first dose; Test type: Superiority or Other; Ratio (Treatment/Placebo) = 0.922, 95.00% CI 2-sided [0.686 to 1.239], Standard Error of Mean 0.148
Statistical Analysis 19: Comparison: Combined Placebo vs Cohort 3-SB-681323, 7.5 mg, 4 h; Comparison at 48 h post first dose; Test type: Superiority or Other; Ratio (Treatment/Placebo) = 0.866, 95.00% CI 2-sided [0.583 to 1.287], Standard Error of Mean 0.198
Statistical Analysis 20: Comparison: Combined Placebo vs Cohort 3-SB-681323, 7.5 mg, 4 h; Comparison at 72 h post first dose; Test type: Superiority or Other; Ratio (Treatment/Placebo) = 0.649, 95.00% CI 2-sided [0.444 to 0.950], Standard Error of Mean 0.190
Statistical Analysis 21: Comparison: Combined Placebo vs Cohort 3-SB-681323, 7.5 mg, 4 h; Comparison at 96 h post first dose; Test type: Superiority or Other; Ratio (Treatment/Placebo) = 0.722, 95.00% CI 2-sided [0.457 to 1.140], Standard Error of Mean 0.228
Statistical Analysis 22: Comparison: Combined Placebo vs Cohort 4-SB-681323, 10 mg, 24 h; Comparison at 6 h post first dose; Test type: Superiority or Other; Ratio (Treatment/Placebo) = 0.897, 95.00% CI 2-sided [0.748 to 1.075], Standard Error of Mean 0.091
Statistical Analysis 23: Comparison: Combined Placebo vs Cohort 4-SB-681323, 10 mg, 24 h; Comparison at 12 h post first dose; Test type: Superiority or Other; Ratio (Treatment/Placebo) = 0.887, 95.00% CI 2-sided [0.703 to 1.119], Standard Error of Mean 0.116
Statistical Analysis 24: Comparison: Combined Placebo vs Cohort 4-SB-681323, 10 mg, 24 h; Comparison at 18 h post first dose; Test type: Superiority or Other; Ratio (Treatment/Placebo) = 0.846, 95.00% CI 2-sided [0.638 to 1.123], Standard Error of Mean 0.142
Statistical Analysis 25: Comparison: Combined Placebo vs Cohort 4-SB-681323, 10 mg, 24 h; Comparison at 24 h post first dose; Test type: Superiority or Other; Ratio (Treatment/Placebo) = 0.812, 95.00% CI 2-sided [0.609 to 1.084], Standard Error of Mean 0.145
Statistical Analysis 26: Comparison: Combined Placebo vs Cohort 4-SB-681323, 10 mg, 24 h; Comparison at 48 h post first dose; Test type: Superiority or Other; Ratio (Treatment/Placebo) = 0.580, 95.00% CI 2-sided [0.394 to 0.855], Standard Error of Mean 0.194
Statistical Analysis 27: Comparison: Combined Placebo vs Cohort 4-SB-681323, 10 mg, 24 h; Comparison at 72 h post first dose; Test type: Superiority or Other; Ratio (Treatment/Placebo) = 0.439, 95.00% CI 2-sided [0.301 to 0.639], Standard Error of Mean 0.188
Statistical Analysis 28: Comparison: Combined Placebo vs Cohort 4-SB-681323, 10 mg, 24 h; Comparison at 96 h post first dose; Test type: Superiority or Other; Ratio (Treatment/Placebo) = 0.451, 95.00% CI 2-sided [0.285 to 0.714], Standard Error of Mean 0.230

24. Secondary Outcome: Markers of Endothelial Cell/Neutrophil Interaction: Mean Soluble Tumor Necrosis Factor Receptors-I
Description: Samples were collected at 6, 12, 18, 24, 48, 72 and 96 h since first dose on Day 1. Mean absolute values of soluble tumor necrosis factor receptors-I levels at these specified time points were reported.
Time Frame: 6, 12, 18, 24, 48, 72 and 96 h since first dose on Day 1
Population: PD Population. Only those participants available at the specified time points were analyzed.
Measure: Geometric Mean (95% Confidence Interval); unit: pg/mL
Arm/Group | Combined Placebo | Cohort 1-SB-681323, 3 mg, 4 h | Cohort 2-SB-681323, 7.5 mg, 24 h | Cohort 3-SB-681323, 7.5 mg, 4 h | Cohort 4-SB-681323, 10 mg, 24 h
Number analyzed (Participants) | 20 | 8 | 10 | 16 | 18
pg/mL
  Time Since 1st Dose, 6 h: number analyzed (Participants) | 18 | 7 | 10 | 16 | 18
  Time Since 1st Dose, 6 h | 2457.23 [2129.05 to 2835.99] | 2089.11 [1653.81 to 2639.00] | 2240.84 [1829.96 to 2743.98] | 2046.04 [1748.13 to 2394.72] | 2267.35 [1961.10 to 2621.42]
  Time Since 1st Dose, 12 h: number analyzed (Participants) | 19 | 7 | 10 | 15 | 17
  Time Since 1st Dose, 12 h | 2448.86 [2124.10 to 2823.28] | 2624.12 [2074.37 to 3319.57] | 2358.84 [1923.30 to 2893.02] | 2151.51 [1829.23 to 2530.58] | 1880.20 [1620.96 to 2180.89]
  Time Since 1st Dose, 18 h: number analyzed (Participants) | 19 | 7 | 10 | 15 | 18
  Time Since 1st Dose, 18 h | 2371.29 [2016.83 to 2788.05] | 2561.58 [1960.37 to 3347.18] | 2175.30 [1725.14 to 2742.92] | 2424.70 [2020.77 to 2909.36] | 1958.95 [1659.12 to 2312.96]
  Time Since 1st Dose, 24 h: number analyzed (Participants) | 19 | 7 | 10 | 16 | 17
  Time Since 1st Dose, 24 h | 2548.08 [2198.02 to 2953.89] | 2423.76 [1898.68 to 3094.06] | 2215.77 [1793.02 to 2738.19] | 2420.75 [2053.68 to 2853.44] | 1939.82 [1664.47 to 2260.71]
  Time Since 1st Dose, 48 h: number analyzed (Participants) | 19 | 7 | 9 | 15 | 17
  Time Since 1st Dose, 48 h | 2466.18 [2072.55 to 2934.58] | 2263.01 [1697.90 to 3016.21] | 2814.63 [2181.24 to 3631.93] | 2388.33 [1961.17 to 2908.52] | 1925.54 [1607.47 to 2306.54]
  Time Since 1st Dose, 72 h: number analyzed (Participants) | 17 | 7 | 9 | 15 | 15
  Time Since 1st Dose, 72 h | 2578.17 [2180.51 to 3048.35] | 2609.42 [1987.30 to 3426.29] | 2893.81 [2268.96 to 3690.73] | 2386.32 [1977.80 to 2879.21] | 1721.54 [1445.26 to 2050.62]
  Time Since 1st Dose, 96 h: number analyzed (Participants) | 17 | 7 | 7 | 14 | 13
  Time Since 1st Dose, 96 h | 2436.04 [2035.38 to 2915.58] | 2844.48 [2133.36 to 3792.64] | 3591.89 [2729.54 to 4726.69] | 2992.91 [2441.71 to 3668.54] | 2094.76 [1720.42 to 2550.55]
Statistical Analysis 1: Comparison: Combined Placebo vs Cohort 1-SB-681323, 3 mg, 4 h; Comparison at 6 h post first dose; Test type: Superiority or Other; Ratio (Treatment/Placebo) = 0.850, 95.00% CI 2-sided [0.646 to 1.119], Standard Error of Mean 0.137
Statistical Analysis 2: Comparison: Combined Placebo vs Cohort 1-SB-681323, 3 mg, 4 h; Comparison at 12 h post first dose; Test type: Superiority or Other; Ratio (Treatment/Placebo) = 1.072, 95.00% CI 2-sided [0.814 to 1.411], Standard Error of Mean 0.138
Statistical Analysis 3: Comparison: Combined Placebo vs Cohort 1-SB-681323, 3 mg, 4 h; Comparison at 18 h post first dose; Test type: Superiority or Other; Ratio (Treatment/Placebo) = 1.080, 95.00% CI 2-sided [0.790 to 1.478], Standard Error of Mean 0.157
Statistical Analysis 4: Comparison: Combined Placebo vs Cohort 1-SB-681323, 3 mg, 4 h; Comparison at 24 h post first dose; Test type: Superiority or Other; Ratio (Treatment/Placebo) = 0.951, 95.00% CI 2-sided [0.715 to 1.266], Standard Error of Mean 0.143
Statistical Analysis 5: Comparison: Combined Placebo vs Cohort 1-SB-681323, 3 mg, 4 h; Comparison at 48 h post first dose; Test type: Superiority or Other; Ratio (Treatment/Placebo) = 0.918, 95.00% CI 2-sided [0.655 to 1.285], Standard Error of Mean 0.168
Statistical Analysis 6: Comparison: Combined Placebo vs Cohort 1-SB-681323, 3 mg, 4 h; Comparison at 72 h post first dose; Test type: Superiority or Other; Ratio (Treatment/Placebo) = 1.012, 95.00% CI 2-sided [0.735 to 1.395], Standard Error of Mean 0.160
Statistical Analysis 7: Comparison: Combined Placebo vs Cohort 1-SB-681323, 3 mg, 4 h; Comparison at 96 h post first dose; Test type: Superiority or Other; Ratio (Treatment/Placebo) = 1.168, 95.00% CI 2-sided [0.831 to 1.640], Standard Error of Mean 0.169
Statistical Analysis 8: Comparison: Combined Placebo vs Cohort 2-SB-681323, 7.5 mg, 24 h; Comparison at 6 h post first dose; Test type: Superiority or Other; Ratio (Treatment/Placebo) = 0.912, 95.00% CI 2-sided [0.713 to 1.167], Standard Error of Mean 0.124
Statistical Analysis 9: Comparison: Combined Placebo vs Cohort 2-SB-681323, 7.5 mg, 24 h; Comparison at 12 h post first dose; Test type: Superiority or Other; Ratio (Treatment/Placebo) = 0.963, 95.00% CI 2-sided [0.753 to 1.233], Standard Error of Mean 0.123
Statistical Analysis 10: Comparison: Combined Placebo vs Cohort 2-SB-681323, 7.5 mg, 24 h; Comparison at 18 h post first dose; Test type: Superiority or Other; Ratio (Treatment/Placebo) = 0.917, 95.00% CI 2-sided [0.693 to 1.214], Standard Error of Mean 0.140
Statistical Analysis 11: Comparison: Combined Placebo vs Cohort 2-SB-681323, 7.5 mg, 24 h; Comparison at 24 h post first dose; Test type: Superiority or Other; Ratio (Treatment/Placebo) = 0.870, 95.00% CI 2-sided [0.673 to 1.123], Standard Error of Mean 0.128
Statistical Analysis 12: Comparison: Combined Placebo vs Cohort 2-SB-681323, 7.5 mg, 24 h; Comparison at 48 h post first dose; Test type: Superiority or Other; Ratio (Treatment/Placebo) = 1.141, 95.00% CI 2-sided [0.840 to 1.550], Standard Error of Mean 0.153
Statistical Analysis 13: Comparison: Combined Placebo vs Cohort 2-SB-681323, 7.5 mg, 24 h; Comparison at 72 h post first dose; Test type: Superiority or Other; Ratio (Treatment/Placebo) = 1.122, 95.00% CI 2-sided [0.837 to 1.505], Standard Error of Mean 0.146
Statistical Analysis 14: Comparison: Combined Placebo vs Cohort 2-SB-681323, 7.5 mg, 24 h; Comparison at 96 h post first dose; Test type: Superiority or Other; Ratio (Treatment/Placebo) = 1.474, 95.00% CI 2-sided [1.063 to 2.045], Standard Error of Mean 0.164
Statistical Analysis 15: Comparison: Combined Placebo vs Cohort 3-SB-681323, 7.5 mg, 4 h; Comparison at 6 h post first dose; Test type: Superiority or Other; Ratio (Treatment/Placebo) = 0.833, 95.00% CI 2-sided [0.672 to 1.031], Standard Error of Mean 0.107
Statistical Analysis 16: Comparison: Combined Placebo vs Cohort 3-SB-681323, 7.5 mg, 4 h; Comparison at 12 h post first dose; Test type: Superiority or Other; Ratio (Treatment/Placebo) = 0.879, 95.00% CI 2-sided [0.707 to 1.092], Standard Error of Mean 0.109
Statistical Analysis 17: Comparison: Combined Placebo vs Cohort 3-SB-681323, 7.5 mg, 4 h; Comparison at 18 h post first dose; Test type: Superiority or Other; Ratio (Treatment/Placebo) = 1.023, 95.00% CI 2-sided [0.800 to 1.307], Standard Error of Mean 0.123
Statistical Analysis 18: Comparison: Combined Placebo vs Cohort 3-SB-681323, 7.5 mg, 4 h; Comparison at 24 h post first dose; Test type: Superiority or Other; Ratio (Treatment/Placebo) = 0.950, 95.00% CI 2-sided [0.761 to 1.187], Standard Error of Mean 0.111
Statistical Analysis 19: Comparison: Combined Placebo vs Cohort 3-SB-681323, 7.5 mg, 4 h; Comparison at 48 h post first dose; Test type: Superiority or Other; Ratio (Treatment/Placebo) = 0.968, 95.00% CI 2-sided [0.743 to 1.262], Standard Error of Mean 0.132
Statistical Analysis 20: Comparison: Combined Placebo vs Cohort 3-SB-681323, 7.5 mg, 4 h; Comparison at 72 h post first dose; Test type: Superiority or Other; Ratio (Treatment/Placebo) = 0.926, 95.00% CI 2-sided [0.718 to 1.193], Standard Error of Mean 0.127
Statistical Analysis 21: Comparison: Combined Placebo vs Cohort 3-SB-681323, 7.5 mg, 4 h; Comparison at 96 h post first dose; Test type: Superiority or Other; Ratio (Treatment/Placebo) = 1.229, 95.00% CI 2-sided [0.936 to 1.613], Standard Error of Mean 0.136
Statistical Analysis 22: Comparison: Combined Placebo vs Cohort 4-SB-681323, 10 mg, 24 h; Comparison at 6 h post first dose; Test type: Superiority or Other; Ratio (Treatment/Placebo) = 0.923, 95.00% CI 2-sided [0.753 to 1.131], Standard Error of Mean 0.102
Statistical Analysis 23: Comparison: Combined Placebo vs Cohort 4-SB-681323, 10 mg, 24 h; Comparison at 12 h post first dose; Test type: Superiority or Other; Ratio (Treatment/Placebo) = 0.768, 95.00% CI 2-sided [0.625 to 0.943], Standard Error of Mean 0.103
Statistical Analysis 24: Comparison: Combined Placebo vs Cohort 4-SB-681323, 10 mg, 24 h; Comparison at 18 h post first dose; Test type: Superiority or Other; Ratio (Treatment/Placebo) = 0.826, 95.00% CI 2-sided [0.655 to 1.042], Standard Error of Mean 0.116
Statistical Analysis 25: Comparison: Combined Placebo vs Cohort 4-SB-681323, 10 mg, 24 h; Comparison at 24 h post first dose; Test type: Superiority or Other; Ratio (Treatment/Placebo) = 0.761, 95.00% CI 2-sided [0.615 to 0.942], Standard Error of Mean 0.106
Statistical Analysis 26: Comparison: Combined Placebo vs Cohort 4-SB-681323, 10 mg, 24 h; Comparison at 48 h post first dose; Test type: Superiority or Other; Ratio (Treatment/Placebo) = 0.781, 95% CI 2-sided [0.608 to 1.003], Standard Error of Mean 0.125
Statistical Analysis 27: Comparison: Combined Placebo vs Cohort 4-SB-681323, 10 mg, 24 h; Comparison at 72 h post first dose; Test type: Superiority or Other; Ratio (Treatment/Placebo) = 0.668, 95.00% CI 2-sided [0.524 to 0.851], Standard Error of Mean 0.121
Statistical Analysis 28: Comparison: Combined Placebo vs Cohort 4-SB-681323, 10 mg, 24 h; Comparison at 96 h post first dose; Test type: Other; Ratio (Treatment/Placebo) = 0.860, 95.00% CI 2-sided [0.659 to 1.122], Standard Error of Mean 0.133

25. Secondary Outcome: Markers of Lung Epithelial Cell Injury: Mean Myeloperoxidase (MPO) Levels
Description: Serum samples were collected at 6, 12, 18, 24, 48, 72 and 96 h since first dose on Day 1. Mean absolute values of MPO levels at these specified time points were reported.
Time Frame: 6, 12, 18, 24, 48, 72 and 96 h since first dose on Day 1
Population: PD Population. Only those participants available at the specified time points were analyzed.
Measure: Geometric Mean (95% Confidence Interval); unit: pg/mL
Arm/Group | Combined Placebo | Cohort 1-SB-681323, 3 mg, 4 h | Cohort 2-SB-681323, 7.5 mg, 24 h | Cohort 3-SB-681323, 7.5 mg, 4 h | Cohort 4-SB-681323, 10 mg, 24 h
Number analyzed (Participants) | 20 | 8 | 10 | 16 | 18
pg/mL
  Time Since 1st Dose, 6 h: number analyzed (Participants) | 17 | 7 | 10 | 15 | 18
  Time Since 1st Dose, 6 h | 66792.4 [50163.43 to 88933.88] | 56739.7 [35517.01 to 90643.64] | 63552.3 [43761.86 to 92292.66] | 44668.1 [32839.83 to 60756.75] | 62108.1 [46378.91 to 83171.68]
  Time Since 1st Dose, 12 h: number analyzed (Participants) | 19 | 7 | 9 | 14 | 17
  Time Since 1st Dose, 12 h | 94963.6 [67732.71 to 133142.20] | 49535.7 [27600.02 to 88905.17] | 85693.0 [52298.94 to 140409.90] | 39467.3 [26518.49 to 58739.05] | 61020.7 [41912.35 to 88840.80]
  Time Since 1st Dose, 18 h: number analyzed (Participants) | 18 | 7 | 10 | 13 | 18
  Time Since 1st Dose, 18 h | 84143.5 [61847.22 to 114477.70] | 70714.1 [42068.42 to 118865.60] | 84578.5 [55836.68 to 128115.10] | 64655.1 [44897.15 to 93107.95] | 67290.8 [48679.72 to 93017.32]
  Time Since 1st Dose, 24 h: number analyzed (Participants) | 17 | 7 | 9 | 14 | 18
  Time Since 1st Dose, 24 h | 104225.0 [78979.78 to 137539.60] | 70943.1 [44906.34 to 112075.90] | 112745.0 [78188.58 to 162572.70] | 59336.2 [43636.15 to 80684.97] | 71506.9 [53769.80 to 95094.96]
  Time Since 1st Dose, 48 h: number analyzed (Participants) | 19 | 7 | 9 | 14 | 17
  Time Since 1st Dose, 48 h | 89181.9 [65657.74 to 121134.40] | 47338.7 [27813.57 to 80570.53] | 92324.6 [59313.52 to 143708.00] | 53458.3 [37505.36 to 76196.80] | 78699.2 [55978.77 to 110641.20]
  Time Since 1st Dose, 72 h: number analyzed (Participants) | 15 | 7 | 9 | 13 | 16
  Time Since 1st Dose, 72 h | 79821.0 [57835.74 to 110163.60] | 88493.3 [53136.78 to 147375.70] | 148310.0 [97377.15 to 225884.00] | 61893.0 [43541.25 to 87979.61] | 73578.6 [52720.51 to 102688.80]
  Time Since 1st Dose, 96 h: number analyzed (Participants) | 17 | 7 | 7 | 11 | 13
  Time Since 1st Dose, 96 h | 70263.5 [50596.69 to 97574.74] | 108777.0 [62959.10 to 187936.90] | 78570.3 [47261.98 to 130618.70] | 84008.1 [55950.12 to 126136.80] | 69268.3 [46791.47 to 102542.10]

26. Secondary Outcome: Mean Area Under the Concentration-time Curve From Zero (Pre-dose) to 24 Hours (AUC0-24)
Description: Absolute values of the mean AUC 0-24 of SB-681323 were reported. PK samples were collected for cohort 1 and 3 at Day 1 (pre-dose, 4, 4.25, 5, 6, 8, 12, 18h), Day 2 (pre-dose and 4h), Day 3 (0, 4, 24, 48h) and for cohort 2 and 4 at Day 1 (pre-dose), Day (pre-dose), Day 3 (pre-dose, 24h10minutes [min], 24h45min, 27, 34, 40, 80 h since doing on Day 3).
Time Frame: For cohort 1 and 3: Day 1 (pre-dose, 4, 4.25, 5, 6, 8, 12, 18h), Day 2 (pre-dose and 4h), Day 3 (0, 4, 24, 48h). For cohort 2 and 4: Day 1 (pre-dose), Day (pre-dose), Day 3 (pre-dose)
Population: Pharmacokinetic (PK) population was defined as patients in the 'All Subjects' population for whom a pharmacokinetic sample was obtained and analyzed. Note: Due to some placebo patients PK samples being assayed in error, the above PK population definition was adjusted to also exclude any patient receiving Placebo.
Measure: Geometric Mean (95% Confidence Interval); unit: h*ng/mL
Arm/Group | Cohort 1-SB-681323, 3 mg, 4 h | Cohort 2-SB-681323, 7.5 mg, 24 h | Cohort 3-SB-681323, 7.5 mg, 4 h | Cohort 4-SB-681323, 10 mg, 24 h
Number analyzed (Participants) | 9 | 12 | 18 | 18
h*ng/mL
  Day 1: number analyzed (Participants) | 9 | 11 | 18 | 17
  Day 1 | 103.222 [85.306 to 124.902] | 186.326 [156.472 to 221.876] | 178.807 [153.644 to 208.090] | 217.862 [182.558 to 259.993]
  Day 2: number analyzed (Participants) | 8 | 11 | 18 | 17
  Day 2 | 112.199 [92.339 to 136.331] | 207.050 [172.749 to 248.163] | 182.590 [156.946 to 212.425] | 237.549 [197.345 to 285.943]
  Day 3: number analyzed (Participants) | 8 | 11 | 17 | 15
  Day 3 | 106.037 [81.444 to 138.057] | 211.282 [177.858 to 250.988] | 188.895 [160.977 to 221.654] | 230.891 [189.316 to 281.598]

27. Secondary Outcome: Mean Average Concentration (Cavg) of SB-681323
Description: Absolute values of mean Cavg of SB-681323 were reported. PK samples were collected for cohort 1 and 3 at Day 1 (pre-dose, 4, 4.25, 5, 6, 8, 12, 18h), Day 2 (pre-dose and 4h), Day 3 (0, 4, 24, 48h) and for cohort 2 and 4 at Day 1 (pre-dose), Day (pre-dose), Day 3 (pre-dose, 24h 10 min, 24h 45min, 27, 34, 40, 80 h since doing on Day 3).
Time Frame: For cohort 1 and 3: Day 1 (pre-dose, 4, 4.25, 5, 6, 8, 12, 18h), Day 2 (pre-dose and 4h), Day 3 (0, 4, 24, 48h). For cohort 2 and 4: Day 1 (pre-dose), Day (pre-dose), Day 3 (pre-dose, 24h 10minutes [min], 24h 45min, 27, 34, 40, 80 h since doing on Day 3)
Population: PK Population. Only those participants available at the specified time points were analyzed.
Measure: Geometric Mean (95% Confidence Interval); unit: ng/mL
Arm/Group | Cohort 1-SB-681323, 3 mg, 4 h | Cohort 2-SB-681323, 7.5 mg, 24 h | Cohort 3-SB-681323, 7.5 mg, 4 h | Cohort 4-SB-681323, 10 mg, 24 h
Number analyzed (Participants) | 9 | 12 | 18 | 18
ng/mL
  Day 1: number analyzed (Participants) | 9 | 11 | 18 | 17
  Day 1 | 4.301 [3.554 to 5.204] | 7.764 [6.520 to 9.245] | 7.450 [6.402 to 8.670] | 9.078 [7.607 to 10.833]
  Day 2: number analyzed (Participants) | 8 | 11 | 18 | 17
  Day 2 | 4.675 [3.847 to 5.680] | 8.627 [7.198 to 10.340] | 7.608 [6.539 to 8.851] | 9.898 [8.223 to 11.914]
  Day 3: number analyzed (Participants) | 8 | 11 | 17 | 15
  Day 3 | 4.418 [3.393 to 5.752] | 8.803 [7.411 to 10.458] | 7.871 [6.707 to 9.236] | 9.620 [7.888 to 11.733]

28. Secondary Outcome: Maximum Observed Concentration (Cmax) of SB-681323
Description: Absolute values of the Cmax of SB-681323 were reported. PK samples were collected for cohort 1 and 3 at Day 1 (pre-dose, 4, 4.25, 5, 6, 8, 12, 18h), Day 2 (pre-dose and 4h), Day 3 (0, 4, 24, 48h) and for cohort 2 and 4 at Day 1 (pre-dose), Day (pre-dose), Day 3 (pre-dose, 24h 10 min, 24h 45min, 27, 34, 40, 80 h since doing on Day 3).
Time Frame: For cohort 1 and 3: Day 1 (pre-dose, 4, 4.25, 5, 6, 8, 12, 18h), Day 2 (pre-dose and 4h), Day 3 (0, 4, 24, 48h). For cohort 2 and 4: Day 1 (pre-dose), Day (pre-dose), Day 3 (pre-dose, 24h 10 min, 24h 45min, 27, 34, 40, 80 h since doing on Day 3)
Population: PK population. Only those participants available at the specified time points were analyzed.
Measure: Geometric Mean (95% Confidence Interval); unit: ng/mL
Arm/Group | Cohort 1-SB-681323, 3 mg, 4 h | Cohort 2-SB-681323, 7.5 mg, 24 h | Cohort 3-SB-681323, 7.5 mg, 4 h | Cohort 4-SB-681323, 10 mg, 24 h
Number analyzed (Participants) | 9 | 11 | 18 | 17
ng/mL
  Day 1 | 21.238 [18.235 to 24.736] | 8.519 [7.098 to 10.225] | 38.032 [33.317 to 43.415] | 10.044 [8.375 to 12.046]
  Day 2: number analyzed (Participants) | 8 | 11 | 18 | 17
  Day 2 | 22.830 [19.533 to 26.683] | 8.842 [7.377 to 10.599] | 38.697 [33.996 to 44.048] | 10.382 [8.647 to 12.466]
  Day 3: number analyzed (Participants) | 8 | 11 | 17 | 15
  Day 3 | 21.888 [18.670 to 25.661] | 8.990 [7.515 to 10.755] | 39.180 [34.157 to 44.943] | 10.131 [8.273 to 12.407]

ADVERSE EVENTS:
Time Frame: Up to follow up period (Day 7).
Description: All subjects population was used for collection of AEs.
Arm/Group | Combined Placebo | Cohort 1-SB-681323, 3 mg, 4 h | Cohort 2-SB-681323, 7.5 mg, 24 h | Cohort 3-SB-681323, 7.5 mg, 4 h | Cohort 4-SB-681323, 10 mg, 24 h
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/9 | 0/12 | 0/18 | 0/18
Serious Adverse Events (participants affected / at risk) | 1/20 | 1/9 | 1/12 | 4/18 | 0/18
Other Adverse Events (participants affected / at risk) | 18/20 | 7/9 | 10/12 | 16/18 | 14/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Combined Placebo (N=20) | Cohort 1-SB-681323, 3 mg, 4 h (N=9) | Cohort 2-SB-681323, 7.5 mg, 24 h (N=12) | Cohort 3-SB-681323, 7.5 mg, 4 h (N=18) | Cohort 4-SB-681323, 10 mg, 24 h (N=18)
Gastrointestinal anastomotic leak (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Wound dehiscence (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Mental impairment (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Quadriplegia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Mental status changes (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Combined Placebo (N=20) | Cohort 1-SB-681323, 3 mg, 4 h (N=9) | Cohort 2-SB-681323, 7.5 mg, 24 h (N=12) | Cohort 3-SB-681323, 7.5 mg, 4 h (N=18) | Cohort 4-SB-681323, 10 mg, 24 h (N=18)
Feeding disorder (Metabolism and nutrition disorders) | 4 | 1 | 1 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 4 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 2 | 0 | 1 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 2 | 0
Hypovolaemia (Metabolism and nutrition disorders) | 2 | 0 | 2 | 0 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 2
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 6 | 4 | 4 | 1 | 3
Constipation (Gastrointestinal disorders) | 4 | 4 | 0 | 2 | 1
Vomiting (Gastrointestinal disorders) | 4 | 0 | 1 | 0 | 1
Ileus (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Pyrexia (General disorders) | 8 | 1 | 6 | 4 | 1
Oedema peripheral (General disorders) | 0 | 1 | 0 | 0 | 1
Asthenia (General disorders) | 0 | 1 | 0 | 0 | 0
Infusion site bruising (General disorders) | 0 | 1 | 0 | 0 | 0
Infusion site extravasation (General disorders) | 1 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 7 | 2 | 3 | 3 | 3
Hypotension (Vascular disorders) | 3 | 1 | 0 | 1 | 0
Deep vein thrombosis (Vascular disorders) | 2 | 0 | 0 | 0 | 0
Bacterial test positive (Investigations) | 1 | 1 | 0 | 1 | 0
Blood potassium decreased (Investigations) | 0 | 0 | 0 | 1 | 2
Hepatic enzyme increased (Investigations) | 1 | 1 | 1 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 1 | 0 | 1 | 0 | 0
Blood pressure increased (Investigations) | 0 | 0 | 0 | 2 | 0
Haemoglobin decreased (Investigations) | 0 | 0 | 0 | 1 | 1
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 0 | 1 | 0
Blood glucose increased (Investigations) | 0 | 1 | 0 | 0 | 0
Blood phosphorus decreased (Investigations) | 0 | 0 | 0 | 0 | 1
Blood potassium increased (Investigations) | 1 | 0 | 0 | 0 | 0
Electrocardiogram QT prolonged (Investigations) | 1 | 0 | 0 | 0 | 0
Electrocardiogram ST segment depression (Investigations) | 1 | 0 | 0 | 0 | 0
Oxygen saturation decreased (Investigations) | 0 | 0 | 0 | 0 | 1
Prothrombin time prolonged (Investigations) | 0 | 0 | 0 | 0 | 1
Sputum culture positive (Investigations) | 1 | 0 | 0 | 0 | 0
Urine output decreased (Investigations) | 0 | 0 | 0 | 0 | 1
White blood cell count increased (Investigations) | 0 | 0 | 0 | 0 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0 | 1 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 1
Bronchial secretion retention (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Agitation (Psychiatric disorders) | 4 | 0 | 2 | 2 | 2
Anxiety (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0
Delirium (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 1 | 0 | 1
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1 | 1
Bradycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Cardiac failure (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Pericardial effusion (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Supraventricular tachycardia (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Ventricular extrasystoles (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Oliguria (Renal and urinary disorders) | 2 | 0 | 0 | 1 | 0
Renal failure acute (Renal and urinary disorders) | 0 | 0 | 1 | 1 | 0
Urinary retention (Renal and urinary disorders) | 0 | 1 | 0 | 1 | 0
Myoglobinuria (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0
Urinary incontinence (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 1 | 1 | 1 | 1 | 1
Coagulopathy (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 2 | 0 | 0 | 1 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 2 | 0
Bacteraemia (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Pneumococcal sepsis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Pneumonia staphylococcal (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 1 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 2
Convulsion (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Lethargy (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Postoperative respiratory distress (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Hypernatraemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
Metabolic alkalosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Vitamin B complex deficiency (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.